# Genetic Risk Assessment for Cancer Education and Empowerment Project (GRACE)

NCT03326713

November 6<sup>th</sup>, 2024



# NON-INTERVENTIONAL/METHODOLOGICAL RESEARCH PROTOCOL TEMPLATE

(HRP-503b)

#### **STUDY INFORMATION**

Title of Project: The Genetic Risk Assessment for Cancer Education and Empowerment (GRACE) Project

## **Principal Investigator:**

Anita Kinney, PhD

**Rutgers Cancer Institute of New Jersey** 

195 Little Albany Street New Brunswick, NJ 08901 Telephone: (732) 235-8871

Email: anita.kinney@rutgers.edu

**Subinvestigators:** 

Antoinette Stroup, PhD Director, Cancer Surveillance Research Program, Rutgers Cancer Institute

Cancer Epidemiology Services, New Jersey State Cancer Registry, NJDOH

Lisa E. Paddock, PhD, MPH Deputy Director, Cancer Surveillance Research Program, Rutgers Cancer Institute

Cancer Epidemiology Services, New Jersey State Cancer Registry, NJDOH

Jie Li, MPH Research Scientist, Cancer Epidemiology Services, NJSCR, NJDOH

Natalia Herman, MPH Research Teaching Specialist, Cancer Surveillance Research Program, RCINJ

PROTOCOL VERSION NUMBER AND DATE: Version 811/6/2024

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



# **Table of Contents**

Skip To Section: Hold CTRL + Click (Below) To Follow Link in Blue

| 1.0 | Research Design |
|------|-----------------------------------------------------------------------|
| 1.1 | Purpose/Specific Aims |
| 1.2 | Research Significance |
| 1.3 | Research Design and Methods |
| 1.4 | Preliminary Data |
| 1.5 | Sample Size Justification |
| 1.6 | Study Variables |
| 1.7 | Specimen Collection As A Primary Source |
| 1.8 | Interviews, Focus Groups, or Surveys and/or Observations |
| 2.0 | Project Management |
| 2.1 | Research Staff and Qualifications |
| 2.2 | Resources Available |
| 2.3 | Research Sites |
| 3.0 | Multi-Site Research Communication & Coordination |
| 3.1 | Non-Rutgers Research Sites |
| 4.0 | Research Data Source/s |
| 4.1 | <u>Primary Data – Subjects and Specimens</u> |
| 4.2 | Subject Selection and Enrollment Considerations |
| 4.3 | Subject Randomization |
| 4.4 | Secondary Subjects |
| 4.5 | Number of Subjects |
| 4.6 | Consent Procedures |
| 4.7 | Special Consent Populations |
| 4.8 | Economic Burden and/or Compensation |
| 4.9 | Risks and Benefits to Subjects |
| 4.10 | Secondary Data – Record/Chart Reviews, Databases, Tissue Banks, Etc. |
| 4.11 | <u>Chart/Record Review Selection</u> |
| 4.12 | Secondary Specimen Collection |
| 5.0 | Special Considerations |
| 5.1 | Health Insurance Portability and Accountability Act (HIPAA) |
| 5.2 | Family Educational Rights and Privacy Act (FERPA) |
| 5.3 | NJ Access to Medical Research Act |
| 5.4 | Code of Federal Regulations Title 45 Part 46 (Vulnerable Populations) |
| 6.0 | Research Data Protection and Reporting |
| 6.1 | <u>Data Management and Confidentiality</u> |
| 6.2 | <u>Data Security</u> |
| 6.3 | Data and Safety Monitoring |
| 6.4 | Reporting Results |
| 7.0 | Data and/or Specimen Banking |
| 8.0 | Other Approvals/Authorizations |
| 9.0 | <u>Bibliography</u> |

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



#### 1.0 Research Design

#### 1.1 Purpose/Specific Aims

The primary purpose of this study is to compare the effectiveness of a usual care (UC) vs. targeted generic print (TP) vs. tailored telephone counseling and navigation intervention (TCN) on cancer genetic risk assessment (CGRA) uptake at 6 months for hereditary breast and ovarian cancer (HBOC). Secondary purposes are: 1) to compare the effectiveness of a TP vs. a TCN intervention vs. UC on CGRA uptake at 12 months, after removal of key access barriers; 2) to compare uptake of genetic testing for HBOC across the three study arms at 6 and 12 months; 3) to compare cognitive (beliefs, attitudes, and knowledge) and affective (distress, stress, fear) intermediate endpoints among women in the three study arms and explore potential underlying theoretical mediating and moderating mechanisms that will further specify and elucidate significant intervention effects; and 4) to perform an economic evaluation alongside this randomized controlled trial to estimate the cost effectiveness of the two interventions compared to each other and usual care, for uptake of CGRA services from the societal and payer perspectives.

The New Jersey State Cancer Registry (NJSCR) will collaborate with investigators from the state cancer registries of Colorado and New Mexico (Dr. Anita Kinney = overall Principal Investigator) to identify women recently diagnosed with high-risk breast and ovarian cancer. The NJSCR will (a) recruit and consent New Jersey patients who are eligible to participate in the study, and (b) securely send contact and cancer-related information to the overall PI for women who consent so that they can be enrolled onto study by the overall PI. This application is for case ascertainment using the NJCSR.

## A. Objectives

AIM 1: Compare the effectiveness of a TP vs. a TCN intervention vs. UC on CGRA uptake 6 months (primary outcome) after the intervention and at 12 months, after removal of key access barriers.

AIM 2: Compare uptake of genetic testing for HBOC across the three study arms at 6 and 12 months.

AIM 3: Compare cognitive (beliefs, attitudes, and knowledge) and affective (distress, stress, fear) intermediate endpoints among women in the three study arms and explore potential underlying theoretical mediating and moderating mechanisms that will further specify and elucidate significant intervention effects.

AIM 4: Perform an economic evaluation alongside this randomized controlled trial to estimate the cost effectiveness of the two interventions compared to each other and usual care, for uptake of CGRA services from the societal and payer perspectives. This aim provides information about the value of the interventions from both societal and payer perspectives, given a cost per effect measure and the uncertainty surrounding the estimate.

#### B. Hypotheses / Research Question(s)

Primary Hypothesis: Compared to UC, CGRA (genetic counseling) uptake at 6 months (primary outcome) will be highest among women participating in the TCN arm followed by women participating in the TP arm.

1.2 Research Significance (Briefly describe the following in 500 words or less):

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



**HBOC Cancer Risks and Genetic Risk Prediction.** Identification of individuals at increased risk of HBOC is crucial for cancer survivors and their families to benefit from biomedical advances. In 2015, approximately 254,000 new cases of ovarian cancer and female breast cancer were diagnosed in the U.S. Germline mutations in the BRCA1 and BRCA2 genes account for 5-10% of breast cancers and 15% of ovarian cancers. <sup>1-3</sup> This translates to 14,000-

27,000 high-risk cancer survivors who may be impacted by HBOC. Women with inherited HBOC gene mutations who have had breast cancer are at higher risk of ovarian cancer and a second breast cancer (Figure 1), and possibly other cancers.<sup>4</sup>

Technological advances in DNA sequencing have now made it possible to test multiple genes simultaneously using multiplex gene panels.<sup>2,5-18</sup>



■ General Population
■ BRCA Mutation

## **CGRA Personalizes Care and is Recommended for**

**High-Risk Breast and Ovarian Cancer Survivors.** CGRA is an evidence-based strategy that informs medical management options that can improve outcomes. <sup>14,17,19</sup> CGRA involves genetic counseling +/- genetic testing. There is evidence that CGRA by genetic professionals improves accuracy of risk perceptions, enables informed decision making, personalizes care, and does not cause adverse psychological outcomes. <sup>14,16,20-22</sup> National

Figure 2. Management of Hereditary Breast and Ovarian Cancer for Survivors



organizations have issued guidelines recommending CGRA for breast and ovarian cancer survivors who may be at risk for HBOC. 17,20,23,24 CGRA in HBOC survivors impacts public health (Figure 2). 4,17 If a mutation is identified, testing for the known gene mutation can be offered to relatives to determine if they have the cancer predisposition. 20,25

Translation of HBOC Discoveries & Guidelines to Practice Has Been Disappointingly Slow. Genetic counseling, guidelines for referral, and testing for HBOC, have been available for >20 years. However, adoption has been slow. It is estimated that  $\leq$ 50% of high-risk cancer patients receive a CGRA referral from their providers, <35% of these women receive genetic counseling and <10% receive testing. Analy women who receive referrals do not adhere to their provider recommendations. Analysis

## 1.3 Research Design and Methods

This is a retrospective cohort study of women diagnosed with aggressive breast or ovarian cancer in New Jersey, New Mexico, and Colorado. This application covers the work being completed in New Jersey only. The NJSCR will identify women recently diagnosed breast and ovarian cancer who meet the following inclusion/exclusion criteria. (Table 1)

We will not include any of the following special populations:

- Adults unable to consent
- Individuals who are not yet adults (infants, children, teenagers)
- Pregnant women
- Prisoners

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



Table 1: Inclusion / Exclusion Criteria for NJSCR recruitment

| Cancer Type | Inclusion | Exclusion |
|---|---|---|
| Breast Cancer survivors | Hispanic or non-Hispanic | Have had prior genetic counseling or |
| | Female | testing for hereditary breast and/or |
| | 21 years of age or older | ovarian cancer |
| | English or Spanish-speaking | Unable to give informed consent |
| | Breast cancer history = | (incoherent, dementia) |
| | breast cancer at the age or before age 50 | No access to a telephone |
| | OR | In hospice care |
| | triple negative breast cancer at or before | Incarcerated |
| | age 60 OR | Permanent residence outside of NJ |
| | two or more primary breast cancers | Planning on relocating out of NJ within |
| | Primary Cancer dx'ed prior to breast | the next year |
| | cancer is OK | |
| | Primary tumor dx'ed after breast cancer | |
| | is OK | |
| Ovarian Cancer Survivors | Hispanic or non-Hispanic | Have had prior genetic counseling or |
| | Female | testing for hereditary breast and/or |
| | 21 years of age or older | ovarian cancer |
| | English or Spanish-speaking | Unable to give informed consent |
| | History of ovarian, fallopian, or | (incoherent, dementia) |
| | peritoneal cancer diagnosed at any age | No access to a telephone |
| | Primary Cancer dx'ed prior to ovarian | In hospice care |
| | cancer is OK | Incarcerated |
| | Primary tumor dx'ed after ovarian cancer | Permanent residence outside of NJ |
| | is OK | Planning on relocating out of NJ within |
| | | the next year |

#### A. Research procedures:

The NJSCR will conduct patient recruitment following their established Standard Operating Procedures (NJSCR Data Repository #Pro20140000992).

Recently diagnosed cases will be identified by staff at the NJSCR and reviewed by a Certified Tumor Registrar (CTR) for study eligibility (Table 1). We will update address information for the case and the physician of record. Each person will be assigned an arbitrary study ID and imported into the study tracking database "CRIMSON." NJSCR staff will send a letter to the patient's diagnosing physician of record to notify the physician that his/her patient is eligible for participation in the study. Physicians are asked to notify NJSCR if the patient should not be contacted for participation (i.e., deceased). Two weeks after the physician letter is mailed, NJSCR staff will send the eligible patient a packet of study materials, including:

- 1. An introductory letter containing a brief description of the study (English or Spanish), a statement of how the patient was determined to be eligible for inclusion into the study, a statement of how the patient was identified via the NJSCR, and a request for the patient's participation;
- 2. Two copies (one to sign and return, one to keep) of an "agreement to contact" sheet that contains all aspects of informed consent and a location to sign;
- 3. An information sheet that contains all aspects of HIPAA;
- 4. An NJSCR Study FAQ brochure which aims to answer common questions about the NJSCR and study participation; and,

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



5. A postage paid return envelope for the completed Agreement to Contact form.

One week (or five business days) after the initial mailing, staff at the NJSCR will conduct six to eight follow-up phone calls at varying times of the day and different days of the week with at least one evening call made between the hours of 5-8pm and at least one call made on a weekend. Those reached by phone will be given the option to provide a verbal consent to be contacted, which will be recorded in the tracking database. A Spanish-speaking NJSCR staff member will contact individuals who indicated Spanish as a preferred language during patient contact. Additional recruitment packets will be mailed upon patient request or if returned for an incorrect address. NJSCR will track all contact with the patient using the CRIMSON tracking database.

NJSCR contracted with Salt City Research to design a tracking tool for patient contact studies, particularly mail and phone contact, and participant response status. CRIMSON works with SEER\*DMS (NJSCR registry database system) and includes modifiable reports and tracking for mode of contact. Key features of CRIMSON include: (1) enhanced report functions and data collection for key recruitment statistics across all studies; (2) enhanced interoperability with SEER\*DMS to reduce manual entry of data and improve data sharing; (3) improved data integrity, quality, consistency, and collection through implementation of validation tools and triggers, elimination of data redundancies, and execution of auto-fill and auto-coding of key variables to remove manual entry of data whenever possible; and (4) implementation of relational structure of the data system allowing for all studies and associated administrative data to be housed within a single data system.

After consent / "Agreement to Participate", NJSCR staff will transfer data securely for consented individuals to the prime site for enrollment and participation in the study.

Briefly, the prime site will randomize the individuals into one of three study arms. NJSCR will not be involved in the intervention. Women will be randomized to one of three study arms: UC, mailed TP, and TCN delivered by a health education specialist. Group assignment will occur at the end of the baseline interview using a computerized randomized list. The interventions will take place ideally within 2 weeks but no more than 30 days upon completion of the baseline survey. Follow-up surveys will be conducted 1 month (to assess mediation), 6 months, and 12 months after randomization for the UC arm, and 1 month, 6 months, and 12 months after the interventions for TP and TCN arms. During the 6 and 12 month surveys, participants will be asked if they'd like to participate in future research. All survey questions will be stored in the REDCap database. The 3 arms will be compared with regard to uptake of CGRA at 6 months (primary outcome) and 12 months, and secondary outcomes including psychosocial and decision-making factors, CGRA preferences, genetic test uptake at 6 and 12 months, and cost outcomes at 6 and 12 months.

- B. Recruitment in New Jersey will begin in July 2018 once SRB and IRB approvals are received and continue through July 2020. The tasks include SRB approval, IRB approval, case identification, "Agreement to Contact", data analysis, and publications.
  - Overall Study Timeline for the Principal Investigator (Dr. Kinney) once the person is enrolled:
  - The duration of a woman's participation in the study will be approximately 12-13 months depending on study arm.
  - The duration estimated for the investigators to complete the study is approximately 5 years and the estimated time needed to complete primary and secondary analyses that address all the study's aims is about 18 months.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



Month 1-7: Start-up, refine data collection and intervention materials, database creation, train health education specialists, IRB approvals

Month 8-32: Recruit and conduct baseline surveys

Months 8-32: Intervention implementation

Months 7-43: Intermediate and final outcome assessments, data cleaning

Months 44-60: Data analysis, presentations, reports, manuscript preparation and publications, and

submit competitive renewal

## 1.4 Preliminary Data

**Solutions are Needed to Expand Reach and Access, and Reduce HBOC-related Disparities.** Psychoeducational interventions that inform, motivate, and address barriers and facilitators to clinical services are typically more effective in facilitating access to recommended health services. 41,45-49 Evidence shows that patients who are equipped with skills are more likely to follow through with recommended care and have better outcomes at reduced costs. 50,51

For our diverse target population, both print and telephone have been found to be acceptable ways to communicate CGRA information but tailored counseling and navigation vs. targeted print has not been effectively tested in this context.<sup>39,52-54</sup> The purpose of this randomized trial is to test the efficacy compared to usual care in increasing CGRA for HBOC. Cancer registries are in an ideal position to identify and reach large numbers of high-risk cancer survivors who may benefit from risk information that can help them make informed decisions about their health and/or information pertinent to their biological relatives.<sup>55,56</sup>

Each year NJSCR participates in a variety of research studies to use data collected by the NJSCR. Eligible cases are actively being contacted for 10 patient contact studies and 2 additional patient contact studies are in the start-up phases. All are approved by the SRB and IRB. Over the past three years we successfully completed 7 patient contact studies that resulted in several scientific publications. A complete bibliography of successful NJSCR research can be found on our website:

http://www.state.nj.us/health/ces/documents/njscr\_bibliography\_seer\_1980\_2017.pdf

## 1.5 Sample Size Justification

The overall study will require a sample size of 642 participants, as shown below in Figure 1, CONSORT flow diagram. The 642 (214 per arm) high-risk breast and ovarian cancer survivors will be randomized to one of the 3 study arms. Participants will be recruited from both the NM, NJ, and CO cancer registries. In New Jersey, we will contact 7,000 breast and ovarian cancer survivors to obtain 700 consents, expecting that 50% of identified individuals sampled and screened for eligibility will fall under our exclusion criteria or will be ineligible for other reasons, 25-28% will consent, and we will retain 80% over the course of the study. Table 2 shows the number of cases available for contact from the NJSCR.

Based on our experience recruiting through population-based tumor registries there are no anticipated barriers or challenges that will prevent us from reaching our accrual goal and we believe that enrollment will be feasible. Standard methods are used to estimate contact and response rates<sup>113</sup> and these rates are consistent with other studies that used similar population-based sampling and recruitment strategies for health promotion intervention studies in our region (response rates are typically higher for female survivors).<sup>54,57,109,114-116</sup> Based on our calculations and considerable experience recruiting individuals from state cancer registries to epidemiologic and

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



behavioral intervention studies, we are confident that we have a sufficient pool of women who are at increased HBOC risk to recruit into the study. Using data from cancer registries in NJ, NM, and CO, we can estimate the number of potentially eligible living female breast and ovarian cancer survivors who meet the criteria for a referral for CGRA by a credentialed genetic professional.

Table 2: Number of Eligible Women, by cancer type, NJ, annual estimates

| Cancer Type | NJ Annual* No. of<br>Eligible Cases | % Hispanic |
|------------------------|-------------------------------------|------------|
| Ovary | 269 | 10 |
| Fallopian Tube | 21 | <1 |
| Peritoneal | 14 | <1 |
| Breast Early Onset | 1849 | 18 |
| Breast Triple Negative | 425 | 16 |
| Breast 2+ primaries | 1059 | 10 |

New Jersey State Cancer Registry October 25, 2016 analytic file. Processed in December 2017.

<sup>\*</sup>Annual averages are based on counts from the five most recent diagnosis years (2011-2015)



Figure 1: Overall Sample Size and Study Design GRACE Study CONSORT Diagram



PI Name: Kinney

Protocol Title: GRACE Project



#### 1.6 Study Variables

#### A. Independent Variables, Interventions, or Predictor Variables

**Intervention Arms.** Following completion of the baseline survey, participants will be randomly assigned to 1 of 3 study arms: 1) a Usual Care (UC) control arm; 2) a mailed Targeted Print arm (TP); and 3) Tailored Counseling & Navigation (TCN) arm. We hypothesize that the TCN intervention will increase CGRA uptake significantly compared to UC and the TP intervention.

**Arm 1- Usual Care:** A usual care arm is included to assess GGRA uptake in the absence of intervention as well as priming from the surveys for the primary outcome analysis.

**Arm 2- Mailed Targeted Print:** Participants randomized to this arm will be mailed an educational brochure within two weeks of completing the baseline survey. The brochure will be available in English and Spanish. It addresses important evidence-based theoretical targets: CGRA guideline (knowledge), threat appraisal (to validate or raise risk perceptions, HBOC seriousness), response efficacy (benefits and expectations about CGRA), self-efficacy messages (CGRA resources, insurance reimbursement, assistance for those with financial challenges), and possible actions to take (make an appointment and discuss with provider). As described in Section D.1, both the targeted print and tailored intervention materials (described below) were developed using formative community engaged research methods.<sup>119</sup>

Arm 3 - Telephone Counseling & Navigation: Within one month of the baseline survey, a bilingual health education specialists will conduct a 30-45 minute (depending on participant needs) telephone health education and counseling session with women randomized to this arm. The intervention will be offered in English or Spanish, depending on the participant's preference. Because theoretically-based tailored messages are generally more effective than generic messages in producing behavioral change, 91,120 we will individualize the psycho-education and navigation session according to each participant's perceptions of threat and efficacy as derived from the EPPM, 41,100 and according to personal factors such as HBOC and CGRA awareness, family history, cultural factors (e.g., ethnicity, language preference, familism, fatalism, family history), psychological and logistical concerns, knowledge, and barriers to CGRA that arise during the phone call. Prior to the telephone session, participants will receive the same brochure that the TP arm receives. After the phone call, participants will receive a tailored followup letter. It will include images tailored to the individual's age, self-identified ethnicity, and family composition. Health education specialists will enter this into the study database using user-friendly study-specific computer screens similar to our previous work. 41,100 The Michigan Tailoring System (MTS), a publicly available software program, will be used to individually tailor messages and images using demographic, clinical and patient-reported data (http://chcr.umich.edu/mts/) for the letter. This information will be derived from the cancer registry data (age, type of cancer diagnoses) and during the survey or phone call (ethnicity, family history, primary care provider (which may be an oncology specialist), threat and efficacy appraisals, concerns (e.g., family member's risk and/or risk of second cancer, family orientation), top two CGRA facilitators/benefits and top two barriers, and action plan.

Both the health education specialists coaching and tailored letter incorporate evidence-based communication and behavior change approaches designed to raise the participant's perceptions about the threat (to herself and atrisk family members), arouse emotions and manage fear, enhance positive beliefs about CGRA (response efficacy), and increase self-efficacy by addressing barriers, facilitators, and motivation to get CGRA. <sup>39,42,51,121-128</sup> The health education specialist will use a MI style to help participants explore their reasons for getting CGRA, resolve ambivalence/decisional conflict, and develop their own action plans. The outline of the call is summarized in Table 3.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



#### **Table 3. Overview of TCN Arm**

## Step 1: Introduction and Rapport Building.

Step 2: Address HBOC Threat Perceptions. To enhance HBOC risk perception, the health education specialist elicits the women's awareness and thoughts about the CGRA referral guidelines and how these guidelines apply to them. The health education specialist provides information about the participant's personal risk for a HBOC-related second cancer and acknowledges that male and female blood relatives may be at increased cancer risk. Although we anticipate that the vast majority of participants will perceive HBOC as serious, their responses will be used to enhance cognitive processing of information.

Step 3: Address Barriers and Efficacy. The health education specialist elicits the participant's response efficacy beliefs, including risk management options for HBOC. If desired by the participant, the health education specialist describes the CGRA/genetic counseling process; its effectiveness in helping women like them and their blood relatives; and addresses questions, concerns or misconceptions about CGRA (e.g., getting CGRA does not mean one has to have a genetic test). The health education specialist uses the "Importance" Ruler (1 - 10 scale) to elicit participant talk around desire and reasons for CGRA. The health education specialist uses the "Readiness" Ruler (1 - 10 scale) to elicit participant talk around ability, confidence, and commitment to obtain CGRA within the next six months. Throughout the interaction, the health education specialist will utilize a series of open-ended questions to elicit and reinforce the participant's reasons for undergoing CGRA. The health education specialist explores factors that the participant believes would increase priority and/or efficacy to get a CGRA. The health education specialist also elicits and addresses the participant's two most important barriers to getting CGRA and attempts to resolve during the phone call.

**Step 4: Construct an Action Plan.** Using readiness ruler and action planning visual aids, the health education specialist prompts the participant to create a personalized action plan. The health education specialist applies implementation intention principles by encouraging the participant to formulate a plan to obtain a CGRA, to determine what her first step will be, as well as when and how she will execute the plan.

**Step 5: Provide Navigation as Needed.** To further bolster self-efficacy and behavior change, the health education specialist offers further assistance (navigation) to help the patient overcome barriers and asks permission to follow-up with them to provide further help as needed. The dose and follow-up navigation activities will be tracked and analyzed as process variables.

Step 6: Summary, Closing and Follow-up. The health education specialist provides a summary of the participant's self-identified primary reasons for getting CGRA, how to overcome the top two barriers as well as the action plan. The health education specialist asks permission to send a letter to the patient's primary provider letting them know that the participant meets the referral criteria for CGRA according to national guidelines and a copy of the participant's tailored letter. For participants who identify barriers, the health education specialist delineates the next steps and schedules a time to follow-up with the patient by phone. A computer generated tailored letter will be mailed immediately after the phone session that includes the women's personalized action plan.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



#### **B. Dependent Variables or Outcome Measures**

- a) Primary Objective: To compare the effectiveness of a usual care (UC) vs. targeted generic print (TP) vs. tailored telephone counseling and navigation intervention (TCN) on cancer genetic risk assessment (CGRA) uptake at 6 months for hereditary breast and ovarian cancer (HBOC).
  - Primary Endpoint: Medical record verified CGRA uptake at 6 months and at 12 months after removal of key access barriers
- b) Secondary Objective 1: Compare uptake of genetic testing for HBOC across the three study arms at 6 and 12 months
  - Secondary Endpoint 1: Medical record verified genetic testing uptake at 6 and 12 months.
- c) Secondary Objective 2: Compare cognitive (beliefs, attitudes, and knowledge) and affective (distress, stress, fear) intermediate endpoints among women in the three study arms and explore potential underlying theoretical mediating and moderating mechanisms that will further specify and elucidate significant intervention effects
  - Secondary Endpoint 2: Measures of cognitive and affective psychological constructs at 1 and 6 months.
- d) Secondary Objective 3: Perform an economic evaluation alongside this randomized controlled trial to estimate the cost effectiveness of the two interventions compared to each other and usual care, for uptake of CGRA services from the societal and payer perspectives. This aim provides information about the value of the interventions from both societal and payer perspectives, given a cost per effect measure and the uncertainty surrounding the estimate.
  - Secondary Endpoint 3: Cost analysis at 6 and 12 months

## 1.7 Specimen Collection as a Primary Source

Not Applicable

#### 1.8 Interviews, Focus Groups, Surveys, and/or Observations

## A. Administration

#### **NJSCR SITE:**

Recently diagnosed cases will be identified by staff at the NJSCR and reviewed by a Certified Tumor Registrar for study eligibility. We will update address information for the case and the physician of record. Each person will be assigned an arbitrary study ID and imported into the study tracking database "CRIMSON." NJSCR staff will send a letter to the patient's diagnosing physician of record to notify the physician that his/her patient is eligible for participation in the study. Two weeks after the physician letter is mailed, NJSCR staff will send the eligible patient a packet of study materials. One week (or five business days) after the initial mailing, staff at the NJSCR will conduct six to eight follow-up phone calls at varying times of the day and different days of the week. Those reached by phone will be given the option to provide a verbal consent to be contacted, which will be recorded in the tracking database. A Spanish-speaking NJSCR staff member will contact individuals who indicated Spanish as a preferred language during patient contact. NJSCR will track all contact with the patient using the CRIMSON tracking database. After consent / "Agreement to Participate", NJSCR staff will transfer data securely for consented individuals to the prime site for enrollment and participation in the study.

#### PRINCIPAL INVESTIGATOR SITE:

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



All interventions and surveys will be conducted by the Principal Investigator at the prime site. Women will be randomized to one of three study arms: UC, mailed TP, and TCN delivered by a health education specialist. Group assignment will occur at the end of the baseline interview using a computerized randomized list.

#### **Timing and Frequency**

The overall order of events for the study are in Table 4. NJSCR is responsible for recruiting cases.

**Table 4: Study Timeline** 

| Who | Task | Timeline |
|---|---|---|
| NJSCR | Recruitment and Consenting | Start - Up Phase August 2018 |
| PI | Enrollment,<br>Baseline Survey &<br>Randomization | Baseline |
| PI | Intervention | 14-30 days post-<br>baseline |
| PI | Follow up surveys | Arm 1: Usual Care (UC) Arm 2: Targeted Mailed Print (TP) Arm 3: Telephone Counseling & Navigation (TCN) |
| PI | 1 month | 30 d > randomization 30 d > intervention 30 d > intervention |
| PI | 6 months | 180 d > randomization 180 d > intervention 180 d > intervention |
| PI | 12 months | 360 d > randomization 360 d > intervention 360 d > intervention |

#### Location

Case recruitment using the New Jersey State Cancer Registry will occur at the NJSCR Trenton Office (135 East State Street, Trenton, NJ) and the New Brunswick office (120 Albany Street, New Brunswick, NJ)

## Procedures For Audio And Visual Recording

Not applicable

#### Person Identifiers

Staff at the New Jersey State Cancer Registry will identify and contact eligible breast and ovarian cancer survivors following their established Standard Operating Procedures (NJSCR Data Repository #Pro20140000992). If a woman would like to participate in the research study, she will be required to sign an informed consent form / "Agreement to Contact" which will describe all aspects of informed consent, contain information about the HIPAA Privacy Rule, and fully describe study participation. If the woman chooses not to participate, she does not have to return the consent form and if she chooses to participate she can withdraw at any time.

On the consent form / "Agreement to Contact" a woman can give the NJSCR staff permission to release private identifiable information (PII) to the Principal Investigator. The variables that will be needed are: name, all elements of the address at diagnosis and current address, telephone number, demographic variables (i.e., gender, race, age, date of birth, etc.) and cancer-related variables (i.e., date of diagnosis, cancer type, etc.). NJSCR will need to provide these variables to the Principal Investigator so that the woman can be contacted for enrollment, baseline survey, randomization, and interventions.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



To protect personal identifiers, each woman will be assigned an arbitrary identification number and this will be used for communication between research staff. Any PII will be transferred in a secure, encrypted manner. All electronic data will be backed up regularly on a secure server. As aforementioned, the biostatisticians who analyze the data will be blinded to participant's study arm. Data for this study, including PIII, will be stored by NJSCR for 6 years after study completion as required by the Rutgers IRB.

#### **B. Study Instruments**

All recruitment materials, surveys, and intervention materials will be available to participants in English or Spanish, depending on their preference. The TCN session will be conducted in English or Spanish, depending on the participant's preference. Spanish materials will be submitted to the IRB after the English materials have been approved. To further facilitate communication, Spanish speaking participants and study staff may use over the phone translation services.

There will be 4 surveys over the course of the study period (baseline, 1 m, 6m, 12 m) and will include different components as described below. These are developed at the prime site.

**CGRA Decision and Genetic Test Uptake:** Participants who have CGRA within 6 months of the intervention (or baseline survey for UC arm) will be considered "completers" of CGRA for the primary outcome. The primary outcome is medical record verified CGRA delivered by the 6-month follow-up. Those reporting that they had CGRA will be asked to sign a medical release form so that we may verify their self-reported CGRA. This approach is extremely feasible and has been successful in ours'41,134 and others'135,136 prior work. We will track the type of provider (e.g., physician, genetic counselor, etc.) who provided CGRA and document their genetics training via the documentation form. Using the same strategy, we will assess CGRA utilization at 12 months. Through the medical record release signed by patients, self-reported genetic testing (including type of test and test result) will also be medical record verified at 6 and 12 months.

**Sociocultural Factors and Cues to Action:** 1) <u>Sociodemographics</u>: age, gender, education, household income, financial status, marital status, rural-urban community area code, <sup>137</sup> living biological children, and health insurance status, country of origin, years lived in the U.S; 2) Medical history: personal/family history of cancer, cancer stage, heath status, comorbidity index; 3) Acculturation: Short Acculturation Scale; <sup>138</sup> 4) Family and friends social support and encouragement to obtain CGRA; <sup>41,139,140</sup> 5) Family orientation: The Familism Scale; <sup>141</sup> 6) Brief Fatalism Scale; <sup>142,143</sup> 7) Health System Distrust; <sup>144</sup> 8) Receipt of a physician/provider recommendation for CGRA; and 9) Primary health care provider received tailored letter in the TPN arm.

Cognitions/Beliefs: 1) Perceived risk: Distinct items with established predictive validity will assess absolute and comparative risk perceptions about risk of carrying a HBOC gene mutation and family members' risk of HBOC; <sup>39,41,54,145,146</sup> 2) Self-efficacy: items assess women's confidence in their ability to locate CGRA services and obtain such services; <sup>39,100</sup> 3) Response efficacy: beliefs about benefits of CGRA in helping prevent HBOC, managing personal cancer risks, providing important information for family, helping make decisions about genetic testing, and helping cope with risks; <sup>42,126</sup> 4) Subjective Numeracy: validated items from the Subjective Numeracy Scale to assess self-reported numeracy skills; <sup>147,148</sup> 5) Genetic Self Efficacy: items assess women's confidence in their ability to understand genetic information and how it applies to their own health; <sup>149-151</sup> 6) Genetic Information Non-Discrimination Act (GINA) Law Confidence: belief that the GINA law would adequately protect against genetic based discrimination; <sup>152</sup> 7) Decisional conflict associated with the CGRA and gene test decisions will be measured with the SURE Scale; <sup>153,154</sup> 8) Decisional satisfaction about CGRA and gene test decisions will be measured with a 4-item scale <sup>155-157</sup> and 3 additional items that assess how they feel about their

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



CGRA/testing decision in relation to their family; 9) Decision Regret Scale will assess regret related to their decision to have or not have CGRA;<sup>54,158</sup> and 10) Several items will assess CGRA and testing intentions.<sup>126</sup>

**Knowledge:** Items from the National Center for Human Genome Research Knowledge Scale and additional items specific to breast and ovarian cancer survivors and misconceptions concerning CGRA and genetic testing will be used. <sup>159,160</sup> We will also ask participants if they heard about or were referred for CGRA and HBOC genetic testing (e.g., BRCA1/2) prior to being contacted for this study.

**Facilitators and Barriers Regarding CGRA**: Items will be drawn from prior research, including our own work.<sup>39,42,122,126</sup> Barriers at the individual, interpersonal, structural, and system-level will be assessed.<sup>39,42,122</sup> Facilitators include but are not limited to: help from family, desire to reduce risk, and referrals from medical professionals. We will also document the most important barriers and facilitators.

**Health Literacy:** Psychometrically validated items <sup>161,162</sup> from the Short Test of Functional Health Literacy in Adults.

**Emotions:** 1) Fear of HBOC risk (self, family): Affect in Risk Scale; <sup>145,163,164</sup> 2) Cancer Worry Scale; <sup>165,166</sup> 3) Psychological distress: anxiety and depression subscales of the Brief Symptom Inventory, <sup>167-169</sup> Short Perceived Stress Scale; <sup>170,171</sup> 4) Defensive Avoidance <sup>172,173</sup>

**CGRA Mode Preferences:** At the 6-month follow-up, we will elicit their preferred mode of CGRA delivery (telephone, internet (Skype), or in-person) and reason for this preference.

**Reactance to Intervention Materials:** At the 1-month survey, participants will be asked if they received and read the print intervention materials (e.g., brochure, tailored letter, reminder action plan) and had telephone coaching.<sup>53</sup> For those who respond "yes," <sup>53,174-176</sup> open-ended questions will also be included regarding what participants liked and did not like about the materials.

**Future Research:** At the 6 and 12 month surveys, participants will be asked if they are interested in participating in future research.

Cost Data Collection: For the economic assessment, we will collect data on: 1) cost of print materials and mailings; 2) health education specialist time to deliver the intervention and follow-up navigation; 3) participant out-of-pocket and time costs; 4) costs associated with the CGRA and genetic test (BRCA1/2 or gene panel test); and 5) overhead related to the intervention (space, etc.). Time will be valued at US wages rates using data from the US Bureau of Labor Statistics. <sup>177</sup> Some costs will obviously differ by study arm (e.g., telephone/internet charges and time), but other differences may be less obvious. Since we are interested in future replication costs, we will focus on intervention delivery costs, including events and health care use. Briefly, health education specialists will record time and resources used delivering the interventions on participant encounter forms; these forms will be compiled to calculate averages. Participants will asked questions regarding how much time they spent, how much childcare they paid for, and how many miles they traveled for each preventive measure, cancer genetic risk assessment, or genetic test they report getting. We have successfully used these methods previously. <sup>54,178,179</sup>



| Measure | Base-<br>line | 1mo | 6mo | 12mo | Description |
|---|---|---|---|---|---|
| General Health and Clinical<br>Information | х | | | | Heath status, co-morbidity index, information on cancer diagnosis(es) |
| Prophylactic Measures | х | | х | х | Assess uptake of and intention to get mastectomy, mammography, breast MRI, oophorectomy, CA 125, and pelvic ultrasound. Participants will also report on how much time they spent getting each procedure, how much childcare they paid for, and how many miles they had to drive. |
| Psychological Distress <sup>167,168</sup> : BSI anxiety ( $\alpha$ = 0.79-0.81); BSI depression ( $\alpha$ = 0.84085); Short PSS <sup>170,171</sup> ( $\alpha$ = 0.84-0.86) | x | x | x | х | Psychological distress will be assessed using the following: anxiety and depression subscales of the Brief Symptom Inventory; 167,168 Short Perceived Stress Scale. 170,171 |
| Cancer Worry: The McCaul Brief Worry Scale <sup>165,166</sup> ( $\alpha$ = 0.78) | х | x | x | Х | Three items will assess cancer worry using the McCaul Brief Worry Scale <sup>165,166</sup> |
| Fear of HBOC: Affect in Risk Scale <sup>145,164</sup> ( $\alpha$ = 0.94) | х | х | x | | Fear of HBOC will be assessed using 6 items in the Affect in Risk Scale. 145,164 |
| Defensive Avoidance | x | x | x | | Four items assess avoidance in thinking about personal and familial inherited cancer risk. 172,173 |
| Perceived HBOC risk for self and family $^{146,180,181}$ . Perceived threat and efficacy regarding HBOC: Risk Behavior Diagnosis Scale (RBDS) $^{182,183}$ ( $\alpha$ = 0.76-0.92) | x | x | х | | Four items assess perceived HBOC risk for self and family <sup>146,180,181</sup> . Threat and efficacy related to HBOC is assessed using the RBDS which assesses cancer-focused EPPM constructs (perceived risk, response efficacy, self-efficacy, cancer severity). <sup>182,183</sup> |
| HBOC Knowledge: National Center for Human Genome Research Knowledge Scale <sup>160</sup> ( $\alpha$ = 0.74) | x | х | | | HBOC knowledge will be assessed using items from the National Center for Human Genome Research Knowledge Scale. 160 Additional items specific to breast and ovarian cancer survivors 159 have been added, as well as items to assess misconceptions concerning hereditary cancer, CGRA, and genetic testing |

PI Name: Kinney

Protocol Title: GRACE Project



| Family Cancer History | х | | | | Family history of cancer: relative, cancer type, age at diagnosis, etc. |
|---|---|---|---|---|---|
| Prior Access to CGRA and Genetic<br>Testing | x | | | | Will assess whether participants had heard about CGRA and/or were referred for CGRA and HBOC genetic testing (e.g., BRCA1/2) prior to being contacted for this study |
| Physician/Health Care Provider<br>Recommendation and<br>Communication | x | x | x | х | Will assess whether healthcare providers have discussed participant's risk of HBOC and CGRA, and how participants feel discussing CGRA and genetic testing with health care provider. |
| Cancer Genetic Risk Assessment<br>(Genetic Counseling) | | x | х | х | Participants will be asked whether they have had CGRA, the provider who conducted the CGRA, and the provider's genetics training. CGRA will be medical record verified. |
| Cancer Genetic Risk Assessment<br>Intention | х | x | х | х | One item will measure future intention to get cancer genetic risk assessment. In follow up surveys, this will only be asked if participant does not report uptake of CGRA |
| HBOC Genetic Testing Uptake | | x | х | х | Participants will be asked whether they have had HBOC genetic testing, what type of genetic test they had, and the facility where the testing was done. Genetic testing will be medical record verified. |
| HBOC Genetic Testing Intention | х | x | х | х | One item will measure future intention to get genetic testing for HBOC. In follow up surveys, this will only be asked if participant does not report uptake of genetic testing. |
| Decisional conflict for CGRA: SURE Scale $^{153,154}$ ( $\alpha$ = 0.86) | | x | х | x | Decisional conflict associated with the CGRA decision will be measured separately with 4 items using the SURE Scale <sup>153,154</sup> |
| Decisional conflict for HBOC genetic testing: Low Literacy Decisional Conflict Scale (DCS)SURE Scale $^{153,154}$ ( $\alpha$ = 0.86) | | | х | х | Decisional conflict associated with the HBOC gene test decision will be measured separately with 4 items using the SURE SCALE <sup>153,154</sup> |
| Decisional satisfaction with CGRA: Satisfaction with Decision Instrument $^{155,156}$ ( $\alpha$ = 0.90). | | | х | х | Decisional satisfaction will be assessed using the Satisfaction with Decision Instrument. Four questions assess their personal satisfaction with their decision and three additional items assess |

PI Name: Kinney

Protocol Title: GRACE Project



| | | | | | how they feel about their CGRA decision in relation to their family. |
|---|---|---|---|---|---|
| Decision Regret Scale <sup>158</sup> $(\alpha = 0.81 \text{-} 0.92)$ | | | х | х | Five items will ask about regret regarding the decision to have or not have CGRA. 158 |
| CGRA and HBOC Genetic Testing<br>Facilitators <sup>42,126</sup> | x | x | x | х | Facilitators include but are not limited to:<br>help from family, desire to reduce risk of<br>second cancers, and help/referrals from<br>medical professionals. |
| CGRA and HBOC Genetic Testing<br>Barriers <sup>39,42,122</sup> | х | х | х | х | Barriers include but are not limited to: low perceived importance, competing demands, family members' lack of support, travel time, lack of insurance reimbursement. |
| Fatalism (fatalismo) and destiny (destino) <sup>142,143</sup> | х | x | | | Fatalism (fatalismo) and destiny (destino) beliefs will be evaluated with three items. 142,143 |
| Competing Life Concerns <sup>126</sup> | х | х | | | Competing life concerns will be evaluated with three items. 126 |
| GINA Confidence | х | х | | | Assess belief that the Genetic Information Non-Discrimination Act (GINA) law would adequately protect against genetic based discrimination. |
| Health System Distrust Scale <sup>144</sup> | х | | | | Nine items measure one's distrust of the<br>Health Care System. This measure has been<br>psychometrically validated. <sup>144</sup> |
| Health Literacy Screen <sup>161,162</sup> | х | | | | Psychometrically validated items used to asses health literacy in adults. 161,162 |
| Genetic Self Efficacy <sup>151</sup> | х | х | х | | Five items used to assess confidence in ability to understand genetic information and how it applies to personal health and disease risk. <sup>151</sup> |
| Subjective Numeracy <sup>147,148</sup> (α=0.78) | х | | | | Three items used to assess self-reported numeracy skills and preferences. |
| Acculturation: | | | | | Acculturation is assessed by country of |
| Short Acculturation Scale <sup>138</sup> | х | | | | origin, time in the U.S., and language preference (five items from the Short |
| $(\alpha = 0.90)$ | | | | | Acculturation Scale). 138 |

PI Name: Kinney

Protocol Title: GRACE Project



| Social support and encouragement to get CGRA <sup>41,139,140</sup> | | x | x | | Six items assess the extent to which family and friends impact one's intention or ability to get a CGRA for HBOC. The measure was expanded from the 2-item measure of family support <sup>139,140</sup> to assess more aspects of family influence; tangible support, emotional support, and normative influence. |
|---|---|---|---|---|---|
| Family Orientation: The Familism Scale $^{141}$ ( $\alpha$ = 0.87) | x | | | | Family orientation (Familism) assess the relative imporance of self and family where the needs of family are more important and take precedence over the needs of any of the family members. The Familism Scale has been used in several Latino samples. 141,184,185 |
| Sociodemographic | х | | | | Age, gender, ethnicity, education, household income, financial status, marital status, rural-urban community area code, <sup>137</sup> living biological children, employment status. |
| Health Insurance Information | х | | x | х | Health insurance status and changes in insurance |
| CGRA Mode Preferences | | | x | | At the 6-month follow-up, for those who have not had genetic counseling but desire it, we will elicit their preferred mode of CGRA delivery: telephone, internet (Skype), and in-person along with the reason underlying their preference. |
| Reactance to Intervention Evaluation Items adapted from previous work <sup>41,53,173-175</sup> | | x | | | At the one month survey, participants will be asked if they received the print intervention materials and telephone health education specialist coaching from the GRACE Project. 53 For those who responded "yes" to specific materials, a set of 174,175 participants will be asked open-ended questions regarding the materials. Participants will also report how much time they spent reviewing materials and speaking to a cancer education specialist. |
| Cancer Education Specialist Follow<br>Up | | | x | х | Participants will report how long they spoke on the phone during follow up calls with the cancer education specialist. |

PI Name: Kinney

Protocol Title: GRACE Project



| Future online adaptations | х | | | Following intervention, internet usage and willingness to search for genetic service information will be assessed. |
|---|---|---|---|---|
| Cost Data | | х | х | Several items will be used to conduct a cost analysis |

#### 2.0 Project Management

#### 2.1 Research Staff and Qualifications

## **New Jersey State Cancer Registry Staff**

## Antoinette Stroup, PhD, NJSCR Site-Principal Investigator

Dr. Stroup is the Director of the New Jersey State Cancer Registry. As such she will be responsible for oversight of this project at the NJSCR, including sample selection, participant recruitment, data collection and quality control. She will lend her expertise in cancer surveillance, population-based survey research and participate in manuscript writing and presentation of study findings at scientific meetings. As the Director of Cancer Epidemiology Services (CES) and the New Jersey State Cancer Registry (NJSCR) and Principal Investigator of the New Jersey SEER contract, she oversees all administrative and operational aspects of the NJSCR, and manage and oversee all research-related activities (e.g., protocol development, institutional review board compliance, patient contact) through the CES Cancer Research Program. She has over 15 years of experience in population-based cancer surveillance methods and research including prior work at two of the highest performing state cancer registries in the SEER Program.

#### Lisa E. Paddock, MPH, PhD - Program Manager

Dr. Paddock is the Deputy Director of the Cancer Surveillance Research Program, which operates under the direction of the NJSCR Director (Dr. Stroup). Dr. Paddock has nearly 20 years of experience in epidemiologic research and patient contact studies, 15 years of which were spent doing research with the NJSCR data. Dr. Paddock's experience is in outcomes research, with specific training in cancer epidemiology, survey research, and health-related quality of life and she is currently a co-investigator in six patient contact studies where NJSCR-CSRP is recruiting and surveying cases. Dr. Paddock has experience in contacting breast and ovarian cancer survivors for case-control studies that are similar to the work proposed in this application.

#### Jie Li, MPH – Team Lead

Ms. Li is a Masters trained epidemiologist and data analyst who is a Research Scientist in the New Jersey State Cancer Registry – Cancer Surveillance Research Program. In this role, Ms. Li conducts registry-based analytics using data from the New Jersey State Cancer Registry database (SEER\*DMS), and other state and national cancer registry data sources available through SEER\*Stat. She is a member of the Patient Contact Studies Team and the Data Linkage Team and assists in linking cohorts with NJSCR data. Additionally, she assists researchers who would like to use NJSCR data in preparing linkage cohort study protocols and IRB applications, analyzes NJSCR data and develops data reports. Ms. Li has several years of experience successfully leading patient contact studies for the NJSCR, including the CEASAR Study and SEER Willingness to Participate.

#### Natalia L. Herman, MPH - Coordinator

Ms. Herman holds a Master's Degree in Public Health with supplemental training in project management and eight years of experience administering, coordinating, and managing survey research projects. Ms. Herman's expertise is in conducting patient contact studies and surveying patients and studies of various aspects of NJSCR data such as rapid case

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



ascertainment and medical record abstraction. Ms. Herman is the Project Manager for the CRIMSON database, providing operational and functional guidance to staff utilizing the database as well as acting as point of contact for the outside consultant, and internal database administrator in the creation of a web-based version. She will coordinate the day-to-day operations of the patient contact staff and provide training to those who are

## Cynthia G. Nunez, BS – Spanish Interviewer

Ms. Nunez is a Research Teaching Specialist III with the NJSCR-Cancer Surveillance Research Program and is the staff member who can translate and speak Spanish to eligible patients. Ms. Nunez has more than 10 years of experience working with patients and sensitive populations prior to her work at NJSCR-CSRP. Ms. Nunez's primary responsibility is maintaining Scientific Review Board and Institutional Review Board approvals for research studies, coordinating patient contact mailings and patient phone calls, and provides training and mentoring for new staff members.

## **Overall Principal Investigator**

Anita Y. Kinney, PhD, RN, Principal Investigator - Dr. Kinney holds the Carolyn R. Surface Endowed Chair in Population Sciences and is Professor of Epidemiology in the Department of Internal Medicine at the University of New Mexico (UNM) School of Medicine. She is also the Associate Director for Cancer Control and Population Sciences at the UNM Cancer Center. Dr. Kinney has primary responsibility for directing all scientific and administrative activities associated with this project. She works closely with the Senior Program Manager and Project Coordinator, who ensures staff are adequately trained and are meeting study progress benchmarks and day-to-day oversight of study staff data collection activities, recruitment, and retention of participants. Dr. Kinney leads the intervention design and implementation strategy, and works closely with the Senior Program Manager and Project Coordinator to ensure adherence to the study's timeline. She will oversee data analysis and dissemination of the study findings and submission of the competitive grant renewal application.

#### 2.2 Resources Available

#### A. Facilities

Cancer cases diagnosed in New Jersey will be obtained from the New Jersey State Cancer Registry (NJSCR), located within the Cancer Epidemiology Services (CES) program at the New Jersey Department of Health (NJDOH). The NJSCR is managed and supported by Rutgers Cancer Institute of New Jersey (CINJ) through a Memorandum of Agreement between the NJ Department of Health and Rutgers, The State University of NJ. NJSCR receives funding from the National Cancer Institute, the Centers for Disease Control, and other state and federal programs. The NJSCR is a population-based cancer registry dedicated to tracking the occurrence of cancer in the state of New Jersey since 1978. The NJSCR contains information on all cancer cases including the type of cancer, race, gender, age residence at diagnosis, first course of treatment, and survival and, has received recognition for its high quality and timely data. The CRP collaborates on and conducts cancer research studies, publishes findings in scientific journals, analyzes data from the NJSCR and produces statewide cancer incidence, mortality and other specialty reports that inform cancer prevention and control efforts.

The NJSCR employs a full complement of experienced cancer registration, research, and information systems personnel to successfully meet its goals for statewide cancer surveillance and research support. Research and data use are primarily managed and conducted by research scientists in the Cancer Surveillance Research Program (CSRP), under the leadership of the Director (Dr. Stroup) and Deputy Director (Dr. Paddock). The senior Research Scientists manage several research studies and participate in cancer control and prevention initiatives using NJSCR data. Investigators are required to work collaboratively with CSRP staff when developing a research protocol using NJSCR data. Staff members at NJSCR and CSRP are well trained in cancer registration and surveillance research

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



including patient contact studies. CES will support this project by providing key technical and research support for patient contact and provide critical content expertise to the research team in regards to cancer surveillance data and interpretation of results.

The physical location of NJSCR: 135 East State Street, 1st Floor, Trenton, NJ 08625 and 120 Albany Street, Tower 2, 8th Floor, New Brunswick, NJ 08903. Location of Data (Hosted by NCI contractors, remotely): Information Management System (IMS), Inc., TierPoint Baltimore Data Center 1401 Russell Street, Baltimore, MD 21230.

Primary registry operations are located at the NJDOH, 135 East State Street, Trenton, NJ 08625 where key card access to the building and registry space on the 1st floor is required. All visitors must be registered with building security. Per state policies, all cancer registry staff must display their state-issued ID at all times while on the premises. (Note: all employees hired through CINJ are issued state IDs upon employment.) Paper-based documents with identifiable data for cancer cases and employees are stored daily at the close of business in locked filing cabinets and drawers. Employees are also required to log- off or lock desktop computers when they step away from their workspace. The registry has staff working at the Rutgers-New Brunswick Campus in CINJ, 120 Albany Street, Tower 2, 8th Floor, where key card access is also required and who follow the same procedures for securing paper-based documents with identifiable information and securing workstations as described above.

## **B. Medical Or Psychological Resources**

Not Applicable

#### C. Research Staff Training

NJSCR staff involved in this study have been with CSRP for up to 5 years, and the majority possess a college or graduate degree. They attend regular trainings for phone interviewing and speaking with cancer survivors regarding NJSCR and study participation. All staff are trained on Confidentiality Procedures and are required to sign a confidentiality agreement annually. Study specific training will include:

- 1. The purpose and scope of the study;
- 2. Review of roles and responsibilities of each staff and NJSCR;
- 3. Review of the questionnaire;
- 4. Review of frequently asking questions.

## 2.3 Research Sites

The NJSCR will facilitate enrollment of New Jersey patients who consent to participate in the study and provide contact information for these consented women to the Principal Investigator so that they can be contacted for study activities. Recruitment of the NJ cases will be performed at the New Jersey State Cancer Registry offices:

- 135 East State Street, 1st Floor, Trenton, NJ 08625
- 120 Albany Street, Tower 2, 8th Floor, New Brunswick, NJ 08903

Recruitment will also occur at the state cancer registries of Colorado and New Mexico, upon IRB approval at the respective site.

## 3.0 Multi-Site Research Communication & Coordination

Not Applicable

## 3.1 Non-Rutgers Site Research

Not Applicable

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



#### 4.0 Research Data Source/s

#### 4.1 Primary Data: Subjects and Specimens

## 4.2 Subject Selection and Enrollment Considerations

A. Recruitment Details – New Jersey State Cancer Registry – Cancer Surveillance Research Program (NJSCR-CSRP) Subjects are recruited through contact by the NJSCR-CSRP, following their established Standard Operating Procedures (NJSCR Data Repository #Pro20140000992).

Recently diagnosed cases will be identified by staff at the NJSCR and reviewed by a Certified Tumor Registrar (CTR) for study eligibility (Table 1). We will update address information for the case and the physician of record. Each person will be assigned an arbitrary study ID and imported into the study tracking database "CRIMSON." NJSCR staff will send a letter to the patient's diagnosing physician of record to notify the physician that his/her patient is eligible for participation in the study. Physicians are asked to notify NJSCR if the patient should not be contacted for participation (i.e., deceased). Two weeks after the physician letter is mailed, NJSCR staff will send the eligible patient a packet of study materials.

One week (or five business days) after the initial mailing, staff at the NJSCR will conduct six to eight follow-up phone calls at varying times of the day and different days of the week with at least one evening call made between the hours of 5-8pm and at least one call made on a weekend. Those reached by phone will be given the option to provide a verbal consent to be contacted, which will be recorded in the tracking database. A Spanish-speaking NJSCR staff member will contact individuals who indicated Spanish as a preferred language during patient contact. Additional recruitment packets will be mailed upon patient request or if returned for an incorrect address. NJSCR will track all contact with the patient using the CRIMSON tracking database.

#### **B. Source of Subjects**

Eligible subjects are sourced directly through the New Jersey State Cancer Registry.

#### C. Method to Identify Potential Subjects

Subjects will be identified from the New Jersey State Cancer Registry using established methods, by a highly trained Research Scientist using the study inclusion criteria below.

#### **D. Subject Screening**

The NJSCR will identify women recently diagnosed breast and ovarian cancer who meet the inclusion/exclusion criteria in Table 1.

- Inclusion Criteria Breast or Ovarian Cancer diagnosis as defined in Table 1.
- Exclusion Criteria Exclusion criteria include not being able to speak or read English, not a resident of New
  Jersey at the time of diagnosis, or currently enrolled in an active patient contact study with NJSCR-CSRP. See
  Table 1.

#### **E. Recruitment Materials**

The eligible patient will be sent a packet of study materials, including:

- 1. An introductory letter containing a brief description of the study (English or Spanish), a statement of how the patient was determined to be eligible for inclusion into the study, a statement of how the patient was identified via the NJSCR, and a request for the patient's participation;
- 2. Two copies (one to sign and return, one to keep) of an "agreement to contact" sheet that contains all aspects of informed consent and a location to sign;

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



- 3. An information sheet that contains all aspects of HIPAA;
- 4. An NJSCR Study FAQ brochure which aims to answer common questions about the NJSCR and study participation; and,
- 5. A postage paid return envelope for the completed Agreement to Contact form.

Materials will be translated to Spanish after English materials are approved.

Lead Site Recruitment Methods – Not Applicable

## 4.3 Subject Randomization

NJSCR will not be involved in the randomization process. Briefly, the Principal Investigator (Dr. Kinney) will randomize consenting women to one of 3 intervention arms using block randomization – (1) Usual care, (2) Mailed Targeted Print, and (3) Telephone Counseling and Navigation. Randomization will be single blinded. Research team members who are assessing the outcomes will be blinded to study arm assignment. Research staff who are conducting follow-up interviews will be blinded to group assignment as much as possible. At the beginning of the follow-up interviews, the interviewer will request that the participant does not reveal the study arm they were assigned to.

#### 4.4 Secondary Subjects

Not Applicable

## 4.5 Number of Subjects

## A. Total Number of Subjects

In New Jersey, we will contact 7,000 breast and ovarian cancer survivors to obtain 700 consents, expecting that 50% of identified individuals sampled and screened for eligibility will fall under our exclusion criteria or will be ineligible for other reasons, 25-28% will consent, and we will retain 80% over the course of the study.

B. Total Number of Subjects If Multicenter Study – Not applicable

#### 4.6 Consent Procedures

#### A. Consent

#### Documenting Consent

NJSCR will obtain consent for contact and document consent using a form and tracking the information in CRIMSON patient tracking database.

- Waiver of <u>Documentation</u> Of Consent Consent will be taken over the telephone by Rutgers Cancer Institute of New Jersey study staff. The subjects will be asked to sign the HIPAA and return it to the CINJ staff members. During COVID 19 they will return the consent form to a staff member with the address included on the return envelope. These HIPAA consent forms will be stored in a locked safe and transferred back to Rutgers CINJ following the COVID 19 pandemic.
- Waiver or Alteration of Consent Process Not Applicable
- Destruction of Identifiers Not Applicable
- Use of Deception/Concealment Not Applicable

#### **B. Consent Process**

#### Location of Consent Process

The consent process will begin by mail for all participants. Participants will receive a recruitment letter announcing the study and inviting participation. The consent to contact contains a brief description of the study. The process will continue at the start of the survey. A consent script will be read to the subject over the phone. All options contain the appropriate contact information if the

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



subject has any questions. If the woman prefers to provide a verbal consent at the time of follow-up, NJSCR will document the verbal consent.

#### Roles for Individuals Involved in Consent

Consent will be obtained by NJSCR staff. The staff has extensive training, supervision, and experience in obtaining consent.

#### Coercion or Undue Influence

All potential subjects are informed that their participation is voluntary. They are also told that any current or future health care will not be affected if they choose not to participate.

## **4.7 Special Consent/Populations**

## A. Minors-Subjects Who Are Not Yet Adults - Not Applicable

- Criteria for Consent of Minors- Not Applicable
- Wards of the State Not Applicable
- Parental/Guardian Permission Not Applicable
- Assent Process Not Applicable

## **B. Non-English Speaking Subjects**

All recruitment materials, surveys, and intervention materials will be available to participants in English or Spanish, depending on their preference. The TCN session will be conducted in English or Spanish, depending on the participant's preference. Spanish materials will be submitted to the IRB after the English materials have been approved. To facilitate communicate between Spanish speaking participants and study staff, participants and study staff may also use over the phone translation services.

#### Process for Non-English Speaking Subjects

The New Jersey State Cancer Registry database indicated Hispanic ethnicity. If a person is Hispanic, then they will receive English and Spanish materials. NJSCR has a Spanish-speaker on staff (Ms. Nunez) who is available to speak with Spanish-speaking subjects for the consent / Agreement to Contact.

## C. Economic Burden and/or Compensation for Subjects

Expenses

There is no cost for participation in the study.

Compensation/Incentives

Compensation will be offered in consideration of the time spent participating in each phase and is estimated to be 45-60 minutes per survey. Participating women will receive a \$50 gift card for each survey that they complete, totaling 4 surveys or \$250.

## D. Risks and Benefits to Subjects

Description of Subject Risk

This study is expected to be of minimal risk to participants. The study involves consent to participate in research studies. The greatest risk involved is the loss of confidentiality. See Provisions to Protect the Privacy Interests of Subjects section below.

- Risks to Non-Subjects Not Applicable
- Minimizing Risks

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



The greatest risk in the study is the loss of privacy. This is minimized using de-identified data (see Provisions to Protect the Privacy Interests of Subjects below).

## Certificate of Confidentiality (CoC) –

To help us protect privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for identifying information. The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). The Certificate of Confidentiality will not be used to prevent disclosure to state or local authorities of harm to self or others.

## Potential Benefits to Subjects

Although the risks to participants are minimal, the personal and familial benefits are that all participants will be provided with education via print material and those in the TPN arm, will receive behavior change counseling and patient navigation. At 6-months, the study will offer to cover the costs of CGRA for all enrolled women across all study arms, should they desire these services.

## Provisions to Protect the Privacy Interests of Subjects

The NJSCR has established policies and procedures governing the use of cancer surveillance data for research including physical access controls, data access controls, and confidentiality and CITI training. On occasion, a cancer patient that has been contacted by the NJSCR for participation in such observational research studies will express concern about his/her cancer diagnosis information being included in the statewide cancer registry. All NJSCR staff are trained in the proper procedures to discuss the statemandated collection of cancer diagnosis information. If the cancer patient expresses discontent over being contacted for inclusion in research studies, the NJSCR staff member will offer the option for the patient to be placed on a "Do Not Contact for Research" list. The patient will no longer be contacted for any research studies.

#### Research Team Access To Subject Data

The NJSCR will obtain consent to be contacted prior to transferring identifiers to the investigators. The NJSCR will extract selected independent variables from the cancer registry for participants that consent to NJSCR. All computers are password protected and in a secure office. The database holding PII is password protected also and is restricted to NJSCR-CSRP research staff. All electronic files are saved on a secure, encrypted server. Paper files are secured in locked file cabinets in the locked office.

#### 4.8 Secondary Data - Not Applicable

- A. Chart/Record Review Selection Not Applicable
- **B. Secondary Specimen Collection Not Applicable**

## 5.0 Special Considerations

## 5.1 Health Insurance Portability and Accountability Act (HIPAA)

NJSCR is a non-HIPAA covered entity.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



- 5.2 Family Educational Rights and Privacy Act (FERPA) Not Applicable
- 5.3 NJ Access to Medical Research Act Not Applicable
- 5.4 Code of Federal Regulations Title 45 Part 46 (Vulnerable Populations) Not Applicable

#### 6.0 Research Data Protection and Reporting

#### 6.1 Data Management and Confidentiality

#### A. Data Analysis Plan

Participants will be randomized into the 3 arms using block randomization. Analyses will be conducted with SAS 9.4 and R 3.2 or updated versions. Outcome variables, along with baseline and follow-up (as applicable) demographic, clinical and psychosocial factors described above, will be summarized by study arm using standard descriptive statistics such as means (standard deviations) for continuous variables and tabulations for categorical variables. Although we do not anticipate baseline differences in the distribution of measured factors between the randomly assigned arms, we will assess for statistical differences using appropriate parametric and nonparametric tests. While the specific aims along with the analyses are described below, some of the analytical strategies across the aims are described as follows: 1) The key study outcomes will be reported that account for missing data using multiple imputation and intent-to-treat (ITT) approaches. Multiple imputation under the Missing at Random assumption will be applied using a Markov Chain Monte Carlo method<sup>186</sup> via PROC MI in SAS, given the expected pattern of non-monotonic missing data. A post hoc approach will address the influence of missing not at random (MNAR) and the effect of attrition on outcomes of interest. Sensitivity analyses will be performed to assess alternative multiple imputation techniques upon the extent of MNAR influences. 2) Multiplicity will be adjusted for the primary outcome analysis using the Holm's adjustment procedure, which guarantees strong error control.<sup>187</sup> The SAS MULTTEST procedure will be used with the marginal p-values. For secondary endpoints, no multiplicity adjustment is considered. All tests will be two-sided. The effect sizes and 95% confidence intervals (CIs) of all outcomes using both ITT, per protocol, and multiple imputed data will be reported regardless of statistical significances.

Analytic Plan for Addressing Specific Aims: Aim 1 is to test the hypothesis that compared to UC, medical record verified CGRA uptake at 6 months, as the primary outcome, will be highest among women participating in the TCN arm followed by women participating in the TP arm. The proportion and its 95% confidence interval (CI) of CGRA uptake for each arm will be calculated using Wilson score interval or the exact binomial CI of Clopper and Pearson method, depending on the data skewness or sample sizes at each time and ethnic and geographic subgroups. For the primary outcome analysis, logistic regression modeling will be employed with the main covariate of arm to estimate an odds ratio (OR) along with a 95% CI. As needed, we will report an adjusted OR, controlling for confounding factors. Potential confounds include age in years, cancer diagnosis site (breast, ovarian or both), family cancer history (yes vs. no), at-risk first-degree relatives (yes vs. no), education level (< high school, high school diploma, >= college), household income (low: below the median income vs. high or as appropriate), time since diagnosis (<5 years, 6-10 years, > 10 years), health insurance (yes vs. no), geographic residence (rural vs. urban), state (NM vs. CO), health literacy (continuous or categorical levels), ethnicity (Hispanic vs. Non-Hispanic), primary language (English vs. Spanish); other psychological, sociocultural and demographic factors will be adjusted as needed. We will also compare the 3 study arms with regard to medical record verified CGRA uptake by 12 months (secondary outcome) after offering to cover the costs of CGRA following the 6-month survey for those

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



who desire but did not access CGRA. Evaluation of the incremental effect will be assessed by comparing the difference of the primary outcome between changed intervention arms (UC to TP/TCN; TP to TCN). For those that availed themselves of "free" CGRA provided through the study, we will describe patient preferences by study arm and other factors (e.g., age, ethnicity, residence area, education, income, literacy, psychosocial factors, and language preference). Model selection with multiple variables will be conducted using AIC and BIC approximation criteria, while including theoretically and practically relevant variables. Aim 2 tests whether there are differences across the 3 study arms with regard to uptake of genetic testing for HBOC at 6 and 12 months. Similar to Aim 1, multivariable regression modeling approach will be performed for the binary outcome (genetic testing yes vs. no) with the main covariate of arm and other confounding variables at each time point. Then, generalized linear mixed effects model (GLMM) will be employed for the two time point outcomes, using binomial distribution with logit link function and adjusting for the correlation within the same subjects to estimate the behavior trend over time. Aim 3 compares cognitive and affective intermediate endpoints among women in the 3 study arms and explores potential underlying theoretical mediating and moderating mechanisms that will further specify and elucidate significant 6-month and 12-month intervention effects, if such effects are observed. The study arms will be compared with regard to beliefs (threat and efficacy), informed decision making indicators (knowledge, decisional conflict, and decision regret) and emotional factors (cancer worry and fear). Arm comparisons will be based on differences in least-square mean changes from baseline to 6 months (including values from the 1-month survey) from an analysis of covariance model containing terms for study arm with baseline scores for as a covariate. Structural equation modeling (SEM) for the hypothesized meditational pathways will be conducted with the procedure of CALIS in SAS and the 'sem' package in R. Before the SEM, all variables in the modeling will be centered with means zero. The SEM will focus on (1) specifying structural equation models; (2) interpreting the model fit statistics and estimation results; (3) testing model with the arms; and (4) analyzing direct and indirect effects. Mediators of intervention effects include threat appraisals, response efficacy, self-efficacy, knowledge, recommendation about CGRA measured at one-month post intervention. Several indices will be used to assess the adequacy of overall model fit: Comparative Fit Index, Standardized Root Mean-Square Residual, and Rootmean Square Error-of Approximation. 188 The interventions may not be beneficial for all study participants. Thus, sensitivity/moderation analysis will be done to identify subgroups for which the intervention has or does not have an effect (e.g., age, diagnosis, time since diagnosis, rural/urban, education level, literacy, acculturation, language preference, close at-risk relative, household income, familism, family support of CGRA, provider recommendation, and cost, travel and time barriers). This will provide important information about subgroups who are particularly receptive or resistant to the effect of each intervention.

**Economic Analysis:** Aim 4 will measure the incremental cost of implementing the interventions from a payer and societal perspective. The payer in this case would be the entity responsible for funding the cancer registry considering patient ascertainment and intervention implementation; therefore, we will estimate recruitment costs, intervention development and delivery costs and downstream costs up to 1-year post intervention. The societal perspective in theory includes all goods and services consumed as a result of the intervention, including the payer costs and patient costs: deductibles, copayments, and cost-sharing for direct medical goods and services in addition to direct non-medical goods and services such as transportation to appointments, and indirect, or opportunity costs incurred as part of the intervention. We will use micro-costing techniques as recommended by the US Panel on Cost-Effectiveness in Health and Medicine and utilized in our past research on the costs of behavioral interventions. Implementation costs will include labor (e.g., registry and study staff, MI trainer, health education specialists) and non-labor (e.g., printing, mailing, costs of CGRA and genetic tests, telephone

Protocol Number: 2018001350 PI Name: Kinney

Protocol Title: GRACE Project



charges, patient-related travel time). Costs will be grouped as variable and fixed costs. We focus on costs of replicating delivery of the intervention and the immediate down-stream consequences (e.g., obtaining CGRA and genetic testing). Costs will be estimated via direct elicitation from participants and medical records to assign fixed price weights. We consider the following outcomes based on a priori trial specifications: 1) average cost per patient for ascertainment, scheduling, health education specialist-participant interaction time; 2) average cost per CGRA and genetic testing; and 3) average time spent with health education specialist. We will also examine overall health care use (including, visits to genetic professionals and other providers, and genetic testing) by study arm (and covariates as needed) at 6 months and 12 months. The incremental cost-effectiveness of one method over another is derived from using the following formula: Incremental cost-effectiveness  $_A = (C_A - C_B)/(E_A - E_B)$  where  $C_A$ and C<sub>B</sub> refer to average total costs of each alternative and E<sub>A</sub> and E<sub>B</sub> refer to average total effectiveness for each alternative. The resulting incremental cost effectiveness ratio (ICER) calculated for each combination of comparators, TCN, TP, and UC, can be used to assess the value provided by alternative A when compared to alternative B, as it represents the investment required for each additional unit of effect gained. All analyses of cost and effectiveness will be completed on an intent-to-treat basis. Uncertainty in estimates will be tested using probabilistic modeling and sensitivity analysis to assess key drivers of results such as rural/urban residence, cancer type, ethnicity, language preference, age, education, household income and family composition (have at least one living at risk first-degree relative). 191 Uncertainty in the ICER will be evaluated using cost-effectiveness acceptability curve plots. 192

Additional analysis: We will apply the RE-AIM framework to assess reach and effectiveness, implementation and adoption issues overall and by ethnic and geographic subgroup, as well as socioeconomic status and cultural variables (e.g., language, medical mistrust). 193-195 We will describe adherence to the theoretical aspects of the intervention and brief MI using MITI global scores. We will also explore whether process variables (dose and timing of health education specialist-participant interactions, intervention fidelity and intervention reactance measures) influence CGRA uptake at 6 and 12 months. Additionally, implementation issues will be assessed, including health education specialist learning needs and challenges related to counseling and navigation. Content and thematic analysis will be employed to evaluate responses to open-ended questions about barriers and facilitators to CGRA and genetic testing, preferences regarding CGRA and perceptions about the interventions and overall study experience. Two coders (AK & KF) code data and inter-rater reliability will be reported.

#### **B.** Power Analysis

The sample size and power evaluation for the proposed study was based on the primary outcome analysis. Given the study's hypothesis that the TCN intervention will have greater effects over both the UC and TP arm, we believe a minimum 12% difference on CGRA uptake 6 months between any intervention arm would be significant from a public health perspective. <sup>197</sup> We expect no greater than 7% CGRA uptake by 6 months in UC, with at least 12% increments for TP and TCN, respectively. With the adjusted significance level of 0.017 (alpha) for the multiple comparisons using

Holm's correction, 182 participants per study arm will provide 95.7% power to detect a 15% difference in the CGRA uptake 6 months between the UC and TP arms. For the comparison between TP and TCN, 182 patients per arm will provide 84.5% power to detect a 15% difference (19% vs. 34%) at the adjusted 0.025 alpha level using the two-sided Likelihood Ratio test. For the secondary analysis, we expect at least 80% power to assess the interventions' effects on ~10-12% change to 15% differences in genetic testing uptake, and small to medium effect sizes of psychosocial targets between the study arms given the measures' standard deviations since our final

Protocol Number: 2018001350 PI Name: Kinney

Protocol Title: GRACE Project



sample size per arm of 182 exceeds the planned final sample size of 164. Randomizing 548 participants based on 1:1:1 relative sizes ensures > 80% power for all contrasts. Assuming up to 20% attrition after baseline assessment, we will recruit 182 individuals for each arm. The sample size and power was evaluated using PASS13 software. <sup>198</sup> A total of 548 individuals will be required (182 per arm x 3 arms). NJSCR will recruit 700 individuals and the remaining sample size will be obtained from other participating registries.

## C. Securing the Data

All computers are password protected and in a secure office. The database holding PII is password protected also and is restricted to NJSCR-CSRP research staff. To protect personal identifiers, each woman will be assigned an arbitrary identification number and this will be used for communication between research staff. Any PII that is consented to be released will be transferred in a secure, encrypted manner.

All electronic data are saved on a secure, encrypted server and backed up regularly on a secure server. Paper files are secured in locked file cabinets in the locked office.

At the Prime Site, the Principal Investigator (Dr. Kinney) will provide each study participant with a Registry Identifier and Participant Identifier. Data will be linked by these two keys. Names and birthdates (and other PHI) that could be used to identify individuals will not be entered into the main study database. These data will be stored in an excel file which will be kept separate from research data. As aforementioned, the biostatisticians who analyze the data will be blinded to participant's study arm.

Data for this study, including PIII, will be stored by NJSCR for 6 years after study completion as required by the Rutgers IRB.

#### **D. Data Quality Control**

Quality Control – The CRIMSoN patient tracking database will reviewed regularly to assure quality.

#### E. Data Handling

At the New Jersey State Cancer Registry, the Site Principal Investigator (Dr. Stroup) will be responsible for data protection and handling. All data will be stored indefinitely. Only authorized and trained research staff will have access to the data and will be responsible for the transmission of the data. Any PII for consented cases will be shared with the Principal Investigator using Rutgers LiFT, or another large file encryption mechanism.

## 6.2 Data Security

The workflow has been designed to limit access to the link between identifiers and the study ID (see Research Design, section h). Access to data will be limited to study personnel. All computers on which analyses will be conducted will be password protected and will be further protected by the Rutgers firewall and malware protection. All data will be transferred using a secure file transfer system (encrypted file, encrypted email, or secure file transfer protocol). Paper copies of raw data will not be produced. Only aggregate results will be published.

6.3 Data and Safety Monitoring – Not Applicable

#### **6.4 Reporting Results**

A. Sharing of Results with Subjects – Not Applicable

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



## B. Individual Results - Not Applicable

#### C. Aggregate Results

Aggregate results will be published in scientific journals and abstracts will be presented at scientific meetings. Abstracts will be posted on the NJSCR website for the public and participants to read. Participants who request copies of scientific findings will be sent any published journal articles.

#### **D. Professional Reporting**

Investigators will also comply with policies and procedures governing the publication of finding from research utilizing NJSCR data, as well, Dr. Stroup and all co-authors will be given opportunity review any abstract/manuscript prior to its submission or use.

Significant contributions to the field of genetics screening will be reported through:

- Poster and/or oral presentations submitted for professional meetings
- Summarized tables described in manuscripts for submission to professional journals such as Cancer

## 7.0 Data and/or Specimen Banking

- A. Storage Methods Not Applicable
- B. Storage Data Not Applicable
- C. Releasing Data/Specimens Not Applicable

## 8.0 Other Approvals/Authorizations

This study has approval by the University of New Mexico Comprehensive Cancer Center and the Colorado Central Cancer Registry as collaborating sites.

## 9.0 Bibliography

- 1. Chen S, Parmigiani G. Meta-analysis of BRCA1 and BRCA2 penetrance. J Clin Oncol. 2007;25(11):1329-1333.
- 2. Bradbury AR, Patrick-Miller L, Domchek S. Multiplex genetic testing: reconsidering utility and informed consent in the era of next-generation sequencing. *Genetics in Medicine*. 2015;17(2):97-98.
- 3. Walker JL, Powell CB, Chen LM, et al. Society of Gynecologic Oncology recommendations for the prevention of ovarian cancer. *Cancer*. 2015.
- 4. Pal T, Vadaparampil ST. Genetic Risk Assessments in Individuals at High Risk for Inherited Breast Cancer in the Breast Oncology Care Setting. *Cancer Control.* 2012;19(4):255-266.
- 5. Domchek SM, Bradbury A, Garber JE, Offit K, Robson ME. Multiplex genetic testing for cancer susceptibility: out on the high wire without a net? 2013;31(10):1267-1270.
- 6. Bradbury AR, Patrick-Miller L, Long J, et al. Development of a tiered and binned genetic counseling model for informed consent in the era of multiplex testing for cancer susceptibility. *Genetics in Medicine*. 2015;17(6):485-492.
- 7. Maxwell KN, Wubbenhorst B, D'Andrea K, et al. Prevalence of mutations in a panel of breast cancer susceptibility genes in BRCA1/2-negative patients with early-onset breast cancer. *Genet Med.* 2015;17(8):630-638.
- 8. Kuchenbaecker KB, Ramus SJ, Tyrer J, et al. Identification of six new susceptibility loci for invasive epithelial ovarian cancer. *Nature genetics*. 2015;47(2):164-171.
- 9. Easton DF, Pharoah PD, Antoniou AC, et al. Gene-panel sequencing and the prediction of breast-cancer risk. *N Engl J Med.* 2015;372(23):2243-2257.
- 10. Minion LE, Dolinsky JS, Chase DM, Dunlop CL, Chao EC, Monk BJ. Hereditary predisposition to ovarian cancer, looking beyond BRCA1/BRCA2. *Gynecologic oncology*. 2015;137(1):86-92.
- 11. Collins FS, Varmus H. A new initiative on precision medicine. *N Engl J Med.* 2015;372(9):793-795.

Protocol Number: 2018001350

PI Name: Kinney

Protocol Title: GRACE Project



- 12. Couch FJ, Hart SN, Sharma P, et al. Inherited mutations in 17 breast cancer susceptibility genes among a large triple-negative breast cancer cohort unselected for family history of breast cancer. 2015;33(4):304-311.
- 13. Slavin TP, Niell-Swiller M, Solomon I, et al. Clinical Application of Multigene Panels: Challenges of Next-Generation Counseling and Cancer Risk Management. *Frontiers in oncology.* 2015;5:208.
- 14. Nelson HD, Pappas M, Zakher B, Mitchell JP, Okinaka-Hu L, Fu R. Risk assessment, genetic counseling, and genetic testing for BRCA-related cancer in women: a systematic review to update the U.S. Preventive Services Task Force recommendation. *Annals of internal medicine*. 2014;160(4):255-266.
- 15. <a href="http://napbc-breast.org/standards/2013standardsmanual.pdf">http://napbc-breast.org/standards/2013standardsmanual.pdf</a>. NAPfBC. Genetic Evaluation and Management 2014, December 2015.
- 16. Radford C, Prince A, Lewis K, Pal T. Factors which impact the delivery of genetic risk assessment services focused on inherited cancer genomics: expanding the role and reach of certified genetics professionals. *Journal of genetic counseling*. 2014;23(4):522-530.
- 17. Robson ME, Bradbury AR, Arun B, et al. American Society of Clinical Oncology Policy Statement Update: Genetic and Genomic Testing for Cancer Susceptibility. 2015;33(31):3660-3667.
- 18. Hiraki S, Rinella ES, Schnabel F, Oratz R, Ostrer H. Cancer risk assessment using genetic panel testing: considerations for clinical application. *Journal of genetic counseling*. 2014;23(4):604-617.
- 19. Domchek SM, Friebel TM, Singer CF, et al. Association of risk-reducing surgery in BRCA1 or BRCA2 mutation carriers with cancer risk and mortality. *Jama-J Am Med Assoc.* 2010;304(9):967-975.
- 20. Daly MB, Pilarski R, Axilbund JE, et al. Genetic/familial high-risk assessment: breast and ovarian, version 1.2014. *Journal of the National Comprehensive Cancer Network : JNCCN.* 2014;12(9):1326-1338.
- 21. Mavaddat N, Peock S, Frost D, et al. Cancer risks for BRCA1 and BRCA2 mutation carriers: results from prospective analysis of EMBRACE. *J Natl Cancer Inst*. 2013;105(11):812-822.
- 22. Cragun D, Pal T. Identification, Evaluation, and Treatment of Patients with Hereditary Cancer Risk within the United States. *ISRN Oncol.* 2013;2013:260847.
- 23. Runowicz CD, Leach CR, Henry NL, et al. American Cancer Society/American Society of Clinical Oncology Breast Cancer Survivorship Care Guideline. 2015.
- 24. Lokich E, Stuckey A, Raker C, Wilbur JS, Laprise J, Gass J. Preoperative genetic testing affects surgical decision making in breast cancer patients. *Gynecologic oncology*. 2014;134(2):326-330.
- 25. Finch A, Wang M, Fine A, et al. Genetic testing for BRCA1 and BRCA2 in the Province of Ontario. *Clinical genetics*. 2015.
- Armstrong J, Toscano M, Kotchko N, et al. Utilization and Outcomes of BRCA Genetic Testing and Counseling in a National Commercially Insured Population: The ABOUT Study. *JAMA oncology*. 2015;1(9):1251-1260.
- 27. Drohan B, Roche CA, Cusack JC, Hughes KS. Hereditary Breast and Ovarian Cancer and Other Hereditary Syndromes: Using Technology to Identify Carriers. *Ann Surg Oncol.* 2012;19(6):1732-1737.
- 28. Febbraro T, Robison K, Wilbur JS, et al. Adherence patterns to National Comprehensive Cancer Network (NCCN) guidelines for referral to cancer genetic professionals. *Gynecologic oncology.* 2015;138(1):109-114.
- 29. Levy DE, Garber JE, Shields AE. Guidelines for Genetic Risk Assessment of Hereditary Breast and Ovarian Cancer: Early Disagreements and Low Utilization. *J Gen Intern Med.* 2009;24(7):822-828.
- 30. Powell CB, Littell R, Hoodfar E, Sinclair F, Pressman A. Does the diagnosis of breast or ovarian cancer trigger referral to genetic counseling? *Int J Gynecol Cancer*. 2013;23(3):431-436.
- 31. Trivers KF, Baldwin LM, Miller JW, et al. Reported referral for genetic counseling or BRCA 1/2 testing among United States physicians. *Cancer*. 2011;117(23):5334-5343.
- 32. Vanstone M, Chow W, Lester L, Ainsworth P, Nisker J, Brackstone M. Recognizing BRCA gene mutation risk subsequent to breast cancer diagnosis in southwestern Ontario. *Can Fam Physician*. 2012;58(5):E258-E266.

PI Name: Kinney

Protocol Title: GRACE Project



- 33. Wood ME, Kadlubek P, Pham TH, et al. Quality of cancer family history and referral for Genetic Counseling and Testing Among Oncology Practices: A Pilot Test of Quality Measures As Part of the American Society of Clinical Oncology Quality Oncology Practice Initiative. *J Clin Oncol.* 2014;32(8):824-829.
- 34. Cragun D, Bonner D, Kim J, et al. Factors associated with genetic counseling and BRCA testing in a population-based sample of young Black women with breast cancer. *Breast Cancer Res Treat*. 2015;151(1):169-176.
- 35. Weitzel JN, Clague J, Martir-Negron A, et al. Prevalence and Type of BRCA Mutations in Hispanics Undergoing Genetic Cancer Risk Assessment in the Southwestern United States: A Report From the Clinical Cancer Genetics Community Research Network. *J Clin Oncol.* 2013;31(2):210-216.
- 36. D'Agincourt-Canning L. Genetic testing for hereditary cancer: challenges to ethical care in rural and remote communities. *HEC forum*: an interdisciplinary journal on hospitals' ethical and legal issues. 2004;16(4):222-233.
- 37. Levy DE, Byfield SD, Comstock CB, et al. Underutilization of BRCA1/2 testing to guide breast cancer treatment: Black and Hispanic women particularly at risk. *Genetics in Medicine*. 2011;13(4):349-355.
- 38. Riesgraf RJ, Veach PM, MacFarlane IM, Leroy BS. Perceptions and Attitudes About Genetic Counseling Among Residents of a Midwestern Rural Area. *J Genet Couns*. 2015;24(4):565-579.
- 39. Gammon AD, Rothwell E, Simmons R, et al. Awareness and Preferences Regarding BRCA1/2 Genetic Counseling and Testing Among Latinas and Non-Latina White Women at Increased Risk for Hereditary Breast and Ovarian Cancer. *J Genet Couns*. 2011;20(6):625-638.
- 40. Cragun D, DeBate RD, Pal T. Applying public health screening criteria: how does universal newborn screening compare to universal tumor screening for Lynch syndrome in adults with colorectal cancer? *Journal of genetic counseling*. 2015;24(3):409-420.
- 41. Kinney AY, Boonyasiriwat W, Walters ST, et al. Telehealth Personalized Cancer Risk Communication to Motivate Colonoscopy in Relatives of Patients With Colorectal Cancer: The Family CARE Randomized Controlled Trial. *J Clin Oncol.* 2014;32(7):654-+.
- 42. Anderson B, McLosky J, Wasilevich E, Lyon-Callo S, Duquette D, Copeland G. Barriers and Facilitators for Utilization of Genetic Counseling and Risk Assessment Services in Young Female Breast Cancer Survivors. *Journal of Cancer Epidemiology*. 2012;2012:11.
- 43. Komenaka IK, Nodora JN, Madlensky L, et al. Participation of low-income women in genetic cancer risk assessment and BRCA 1/2 testing: the experience of a safety-net institution. *J Community Genet*. 2015.
- 44. van Riel E, van Dulmen S, Ausems MG. Who is being referred to cancer genetic counseling? Characteristics of counselees and their referral. *J Community Genet*. 2012;3(4):265-274.
- 45. Sabatino SA, Lawrence B, Elder R, et al. Effectiveness of interventions to increase screening for breast, cervical, and colorectal cancers: nine updated systematic reviews for the guide to community preventive services.

  American journal of preventive medicine. 2012;43(1):97-118.
- 46. Marcus AC, Diefenbach MA, Stanton AL, et al. Cancer patient and survivor research from the cancer information service research consortium: a preview of three large randomized trials and initial lessons learned. *J Health Commun*. 2013;18(5):543-562.
- 47. Myers RE, Bittner-Fagan H, Daskalakis C, et al. A randomized controlled trial of a tailored navigation and a standard intervention in colorectal cancer screening. Cancer epidemiology, biomarkers & prevention: a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology. 2013;22(1):109-117.
- 48. Manne S, Jacobsen PB, Ming ME, Winkel G, Dessureault S, Lessin SR. Tailored versus generic interventions for skin cancer risk reduction for family members of melanoma patients. *Health psychology : official journal of the Division of Health Psychology, American Psychological Association.* 2010;29(6):583-593.
- 49. Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. *Psychol Bull.* 2007;133(4):673-693.

PI Name: Kinney

Protocol Title: GRACE Project



- 50. Simmons LA, Wolever RQ, Bechard EM, Snyderman R. Patient engagement as a risk factor in personalized health care: a systematic review of the literature on chronic disease. *Genome Med.* 2014;6.
- 51. Mays D, Sharff ME, DeMarco TA, et al. Outcomes of a systems-level intervention offering breast cancer risk assessments to low-income underserved women. *Familial Cancer*. 2012;11(3):493-502.
- 52. Peshkin BN, Kelly S, Nusbaum RH, et al. Patient Perceptions of Telephone vs. In-Person BRCA1/BRCA2 Genetic Counseling. *Journal of genetic counseling*. 2015.
- 53. Simmons RG, Walters ST, Pappas LM, et al. Implementation of Best Practices Regarding Treatment Fidelity in the Family Colorectal Cancer Awareness and Risk Education Randomized Controlled Trial. *SAGE Open.* 2014;4(4).
- 54. Kinney AY, Butler KM, Schwartz MD, et al. Expanding Access to BRCA1/2 Genetic Counseling with Telephone Delivery: A Cluster Randomized Trial. *Jnci-J Natl Cancer I.* 2014;106(12).
- 55. Chen VW, Eheman CR, Johnson CJ, et al. Enhancing cancer registry data for comparative effectiveness research (CER) project: overview and methodology. *J Registry Manag.* 2014;41(3):103-112.
- 56. Ryerson AB, Eheman C, Styles T, Rycroft R, Snyder C. Connecting the Dots: Linking the National Program of Cancer Registries and the Needs of Survivors and Clinicians. *American journal of preventive medicine*. 2015;49(6 Suppl 5):S528-535.
- 57. Carpentier MY, Tiro JA, Savas LS, et al. Are cancer registries a viable tool for cancer survivor outreach? A feasibility study. *J Cancer Surviv*. 2013;7(1):155-163.
- 58. Glanz K, Bishop DB. The Role of Behavioral Science Theory in Development and Implementation of Public Health Interventions. *Annu Rev Publ Health.* 2010;31:399-418.
- 59. Riekert KA, Ockene JK, Pbert L. *Handbook of health behavior change.* 4th edition. ed. New York, NY: Springer Publishing Company, LLC; 2014.
- 60. Witte K. Putting the Fear Back into Fear Appeals the Extended Parallel Process Model. *Commun Monogr.* 1992;59(4):329-349.
- 61. Witte K, Allen M. A meta-analysis of fear appeals: Implications for effective public health campaigns. *Health Educ Behav.* 2000;27(5):591-615.
- 62. Schwarzer R. Models of health behaviour change: Intention as mediator or stage as moderator? *Psychol Health.* 2008;23(3):259-262.
- 63. Schwarzer R, Lippke S, Ziegelmann JP. Health action process approach A research agenda at the Freie Universitat Berlin to examine and promote health behavior change. *Z Gesundheitspsychol.* 2008;16(3):157-160.
- 64. O'Connor AM, Jacobsen MJ, Stacey D. An evidence-based approach to managing women's decisional conflict. *J Obstet Gynecol Neonatal Nurs.* 2002;31(5):570-581.
- 65. Rogers R. Cognitive and physiological processes in fear appeals and attitude change: A Revised theory of protection motivation. In: Cacioppo J, Petty, R., ed. *Social Psychophysiology*. New York, NY: Guilford Press; 1983.
- 66. Ajzen I. The theory of planned behaviour: reactions and reflections. *Psychol Health*. 2011;26(9):1113-1127.
- 67. Fishbein M, Ajzen I. Theory-based behavior change interventions: comments on Hobbis and Sutton. *Journal of health psychology.* 2005;10(1):27-31; discussion 37-43.
- 68. Becker MH, Janz NK. Behavioral science perspectives on health hazard/health risk appraisal. *Health Services Research*. 1987;22(4):537-551.
- 69. Janz NK, Becker MH. The Health Belief Model: a decade later. Health Educ Q. 1984;11(1):1-47.
- 70. Sampson J, Witte K, Morrison K, Liu WY, Hubbell AP, Murray-Johnson L. Addressing cultural orientations in fear appeals: promoting AIDS-protective behaviors among Mexican immigrant and African American adolescents and American and Taiwanese college students. *J Health Commun.* 2001;6(4):335-358.
- 71. Maloney E, Lapinski, MK and Witte K. Fear Appeals and Persuasion: A Review and Update of the Extended Parallel Process Model. *Social and Personality Psychology Compass.* 2011;5:206-219.
- 72. Gollwitzer PM. Implementation intentions Strong effects of simple plans. *Am Psychol.* 1999;54(7):493-503.

PI Name: Kinney

Protocol Title: GRACE Project



- 73. Kwasnicka D, Presseau J, White M, Sniehotta FF. Does planning how to cope with anticipated barriers facilitate health-related behaviour change? A systematic review. *Health Psychol Rev.* 2013;7(2):129-145.
- 74. Schwarzer R. Self-regulatory Processes in the Adoption and Maintenance of Health Behaviors. *Journal of health psychology.* 1999;4(2):115-127.
- 75. Sheeran P. Intention-behavior relations: A conceptual and empirical review *European Review of Social Psychology.* 2002;12:1-36.
- 76. Quality AfHRa. Decision Aids for Cancer Screening and Treatment Comparative Effectiveness Review Number 145. In: Services USDoHaH, ed. Vol AHRQ Publication No. 15-EHC002-EF. Rockville, Maryland2014.
- 77. The Guide to Community Preventive Services. The Community Guide. What Works to Promote Health. Increasing Cancer Screening: Small Media Targeting Clients. <a href="http://www.thecommunityguide.org/index.html">http://www.thecommunityguide.org/index.html</a>. Accessed Dec. 2, 2015.
- 78. Research-tested Intervention Programs (RTIPs). http://rtips.cancer.gov/rtips/index.do. Accessed Dec. 2, 2015.
- 79. Muusses LD, van Weert JCM, van Dulmen S, Jansen J. Chemotherapy and information-seeking behaviour: characteristics of patients using mass-media information sources. *Psycho-Oncology*. 2012;21(9):993-1002.
- 80. Talosig-Garcia M, Davis SW. Information-seeking behavior of minority breast cancer patients: an exploratory study. *J Health Commun.* 2005;10 Suppl 1:53-64.
- 81. Walsh JM, Salazar R, Nguyen TT, et al. Healthy colon, healthy life: a novel colorectal cancer screening intervention. *American journal of preventive medicine*. 2010;39(1):1-14.
- 82. Bastani R, Glenn BA, Maxwell AE, et al. Randomized trial to increase colorectal cancer screening in an ethnically diverse sample of first-degree relatives. *Cancer*. 2015;121(17):2951-2959.
- 83. Hawkins RP, Kreuter M, Resnicow K, Fishbein M, Dijkstra A. Understanding tailoring in communicating about health. *Health Educ Res.* 2008;23(3):454-466.
- 84. Kreuter MW, Wray RJ. Tailored and targeted health communication: strategies for enhancing information relevance. *Am J Health Behav.* 2003;27 Suppl 3:S227-232.
- 85. Sanders Thompson VL, Cavazos-Rehg PA, Jupka K, et al. Evidential preferences: cultural appropriateness strategies in health communications. *Health Educ Res.* 2008;23(3):549-559.
- 86. Glanz K, Escoffery C, Elliott T, Nehl EJ. Randomized Trial of Two Dissemination Strategies for a Skin Cancer Prevention Program in Aquatic Settings. *Am J Public Health*. 2015;105(7):1415-1423.
- 87. Glanz K, Volpicelli K, Jepson C, Ming ME, Schuchter LM, Armstrong K. Effects of tailored risk communications for skin cancer prevention and detection: the PennSCAPE randomized trial. *Cancer epidemiology, biomarkers & prevention: a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology.* 2015;24(2):415-421.
- 88. McBride CM, Birmingham WC, Kinney AY. Health psychology and translational genomic research: bringing innovation to cancer-related behavioral interventions. *Am Psychol.* 2015;70(2):91-104.
- 89. Kreuter MW, Strecher VJ, Glassman B. One size does not fit all: the case for tailoring print materials. *Ann Behav Med.* 1999;21(4):276-283.
- 90. Miller SM, Hui SK, Wen KY, et al. Tailored telephone counseling to improve adherence to follow-up regimens after an abnormal pap smear among minority, underserved women. *Patient Educ Couns.* 2013;93(3):488-495.
- 91. Steffen LE, Boucher KM, Damron BH, et al. Efficacy of a Telehealth Intervention on Colonoscopy Uptake When Cost Is a Barrier: The Family CARE Cluster Randomized Controlled Trial. *Cancer Epidem Biomar.* 2015;24(9):1311-1318.
- 92. Katz ML, Fisher JL, Fleming K, Paskett ED. Patient activation increases colorectal cancer screening rates: a randomized trial among low-income minority patients. *Cancer epidemiology, biomarkers & prevention : a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology.* 2012;21(1):45-52.

PI Name: Kinney

Protocol Title: GRACE Project



- 93. Singal AG, Gupta S, Tiro JA, et al. Outreach invitations for FIT and colonoscopy improve colorectal cancer screening rates: A randomized controlled trial in a safety-net health system. *Cancer.* 2015.
- 94. Glick SB, Clarke AR, Blanchard A, Whitaker AK. Cervical cancer screening, diagnosis and treatment interventions for racial and ethnic minorities: a systematic review. *J Gen Intern Med.* 2012;27(8):1016-1032.
- 95. Glanz K, Rimer BK, Viswanath K. *Health behavior and health education : theory, research, and practice.* 4th ed. San Francisco, CA: Jossey-Bass; 2008.
- 96. Medicine) IIo. Clinical Practice Guidelines We Can Trust. Washington, D.C.: The National Academies Press;2011.
- 97. Paskett ED, Harrop JP, Wells KJ. Patient navigation: an update on the state of the science. *CA Cancer J Clin.* 2011;61(4):237-249.
- 98. Miller WR, Rollnick S. *Motivational interviewing : helping people change.* 3rd ed. New York, NY: Guilford Press; 2013.
- 99. Miller WR, Rollnick S. The effectiveness and ineffectiveness of complex behavioral interventions: impact of treatment fidelity. *Contemp Clin Trials*. 2014;37(2):234-241.
- 100. Pengchit W, Walters ST, Simmons RG, et al. Motivation-based intervention to promote colonoscopy screening: an integration of a fear management model and motivational interviewing. *Journal of health psychology*. 2011;16(8):1187-1197.
- 101. Hall K, Gibbie T, Lubman DI. Motivational interviewing techniques facilitating behaviour change in the general practice setting. *Aust Fam Physician*. 2012;41(9):660-667.
- Hall K, Staiger PK, Simpson A, Best D, Lubman DI. After 30 years of dissemination, have we achieved sustained practice change in motivational interviewing? *Addiction*. 2015.
- 103. Schwalbe CS, Oh HY, Zweben A. Sustaining motivational interviewing: a meta-analysis of training studies. *Addiction*. 2014;109(8):1287-1294.
- 104. Miller WR, Rose GS. Toward a theory of motivational interviewing. *Am Psychol.* 2009;64(6):527-537.
- 105. Miller WR, Rose GS. Motivational interviewing and decisional balance: contrasting responses to client ambivalence. *Behav Cogn Psychother*. 2015;43(2):129-141.
- 106. Corsino L, Rocha-Goldberg MP, Batch BC, Ortiz-Melo DI, Bosworth HB, Svetkey LP. The Latino Health Project: Pilot Testing a Culturally Adapted Behavioral Weight Loss Intervention in Obese and Overweight Latino Adults. *Ethnic Dis.* 2012;22(1):51-57.
- 107. Rocha-Goldberg MD, Corsino L, Batch B, et al. Hypertension Improvement Project (HIP) Latino: results of a pilot study of lifestyle intervention for lowering blood pressure in Latino adults. *Ethnic Health*. 2010;15(3):269-282.
- 108. Connor AE, Baumgartner RN, Baumgartner KB, et al. Associations between ALOX, COX, and CRP polymorphisms and breast cancer among Hispanic and non-Hispanic white women: The breast cancer health disparities study. *Mol Carcinogen*. 2015;54(12):1541-1553.
- 109. Hill DA, Horick NK, Isaacs C, et al. Long-term risk of medical conditions associated with breast cancer treatment. Breast Cancer Res Treat. 2014;145(1):233-243.
- 110. Lowery JT, Horick N, Kinney AY, et al. A randomized trial to increase colonoscopy screening in members of high-risk families in the colorectal cancer family registry and cancer genetics network. *Cancer epidemiology, biomarkers & prevention : a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology.* 2014;23(4):601-610.
- 111. Slattery ML, Sweeney C, Herrick J, et al. ESR1, AR, body size, and breast cancer risk in Hispanic and non-Hispanic white women living in the Southwestern United States. *Breast Cancer Res Treat*. 2007;105(3):327-335.
- 112. Simmons RG, Lee YC, Stroup AM, et al. Examining the challenges of family recruitment to behavioral intervention trials: factors associated with participation and enrollment in a multi-state colonoscopy intervention trial. *Trials*. 2013;14:116.

PI Name: Kinney

Protocol Title: GRACE Project



- 113. American Association of Public Opinion Research: Response Rates An Overview.

  <a href="http://www.aapor.org/AAPORKentico/Education-Resources/For-Researchers/Poll-Survey-FAQ/Response-Rates-An-Overview.aspx">http://www.aapor.org/AAPORKentico/Education-Resources/For-Researchers/Poll-Survey-FAQ/Response-Rates-An-Overview.aspx</a>. Accessed Dec. 2, 2015.
- 114. Ziogas A, Horick NK, Kinney AY, et al. Clinically relevant changes in family history of cancer over time. *Jama-J Am Med Assoc.* 2011;306(2):172-178.
- 115. Ashing K, Rosales M, Fernandez A. Exploring the influence of demographic and medical characteristics of African-American and Latinas on enrollment in a behavioral intervention study for breast cancer survivors. *Qual Life Res.* 2015;24(2):445-454.
- 116. Ashing K, Rosales M. A telephonic-based trial to reduce depressive symptoms among Latina breast cancer survivors. *Psychooncology*. 2014;23(5):507-515.
- 117. Altman DG, Moher D, Schulz KF. Improving the reporting of randomised trials: the CONSORT Statement and beyond. *Statistics in medicine*. 2012;31(25):2985-2997.
- 118. Moher D, Hopewell S, Schulz KF, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. *International journal of surgery*. 2012;10(1):28-55.
- 119. Doak LG, Doak CC, Meade CD. Strategies to improve cancer education materials. *Oncology nursing forum*. 1996;23(8):1305-1312.
- 120. Edwards AGK, Naik G, Ahmed H, et al. Personalised risk communication for informed decision making about taking screening tests. *Cochrane Db Syst Rev.* 2013(2).
- 121. Ricker C, Lagos V, Feldman N, et al. If we build it ... will they come?--establishing a cancer genetics services clinic for an underserved predominantly Latina cohort. *Journal of genetic counseling*. 2006;15(6):505-514.
- 122. Kinney AY, Gammon A, Coxworth J, Simonsen SE, Arce-Laretta M. Exploring attitudes, beliefs, and communication preferences of Latino community members regarding BRCA1/2 mutation testing and preventive strategies. *Genetics in Medicine*. 2010;12(2):105-115.
- 123. Scherr CL, Vasquez E, Quinn GP, Vadaparampil ST. Genetic Counseling for Hereditary Breast and Ovarian Cancer among Puerto Rican Women Living in the United States. *Reviews on recent clinical trials.* 2015;9(4):245-253.
- 124. Adams I, Christopher J, Williams KP, Sheppard VB. What Black Women Know and Want to Know About Counseling and Testing for BRCA1/2. *J Cancer Educ.* 2015;30(2):344-352.
- 125. Sussner KM, Edwards T, Villagra C, et al. BRCA Genetic Counseling Among At-Risk Latinas in New York City: New Beliefs Shape New Generation. *J Genet Couns*. 2015;24(1):134-148.
- 126. Sussner KM, Jandorf L, Thompson HS, Valdimarsdottir HB. Barriers and facilitators to BRCA genetic counseling among at-risk Latinas in New York City. *Psycho-Oncology*. 2013;22(7):1594-1604.
- 127. Glenn BA, Chawla N, Bastani R. Barriers to Genetic Testing for Breast Cancer Risk among Ethnic Minority Women: An Exploratory Study. *Ethnic Dis.* 2012;22(3):267-273.
- 128. Sussner KM, Edwards TA, Thompson HS, et al. Ethnic, racial and cultural identity and perceived benefits and barriers related to genetic testing for breast cancer among at-risk women of African descent in New York City. *Public health genomics*. 2011;14(6):356-370.
- 129. Bellg AJ, Borrelli B, Resnick B, et al. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. *Health Psychology*. 2004;23(5):443-451.
- 130. Bennett GA, Roberts HA, Vaughan TE, Gibbins JA, Rouse L. Evaluating a method of assessing competence in Motivational Interviewing: a study using simulated patients in the United Kingdom. *Addictive behaviors*. 2007:32(1):69-79.
- 131. Borrelli B. The assessment, monitoring, and enhancement of treatment fidelity in public health clinical trials. *Journal of public health dentistry*. 2011;71 Suppl 1:S52-63.
- Borrelli B, Sepinwall D, Ernst D, et al. A new tool to assess treatment fidelity and evaluation of treatment fidelity across 10 years of health behavior research. *Journal of consulting and clinical psychology.* 2005;73(5):852-860.

PI Name: Kinney

Protocol Title: GRACE Project



- 133. Moyers TM, JK; Ernst, D. *Motivational Interviewing Treatment Integrity Coding Manual 4.1* (*MITI 4.1*). Albuquerque, NM: University of New Mexico;2014.
- 134. Levine FR, Coxworth JE, Stevenson DA, Tuohy T, Burt RW, Kinney AY. Parental Attitudes, Beliefs, and Perceptions about Genetic Testing for FAP and Colorectal Cancer Surveillance in Minors. *J Genet Couns*. 2010;19(3):269-279.
- 135. Cragun D, Camperlengo L, Robinson E, et al. Differences in BRCA counseling and testing practices based on ordering provider type. *Genet Med.* 2015;17(1):51-57.
- 136. Hamann HA, Tiro JA, Sanders JM, et al. Validity of self-reported genetic counseling and genetic testing use among breast cancer survivors. *J Cancer Surviv.* 2013;7(4):624-629.
- 137. University of Washington Rural Health Research Center: Rural-urban commuting area codes (version 2.0) http://depts.washington.edu/uwruca/. Accessed March 30, 2015.
- 138. Marin G, Sabogal F, Marin BV, Otero-Sabogal R, Perez-Stable EJ. Development of a short acculturation scale for Hispanics. *Hispanic Journal of Behavioral Sciences*. 1987;9(2):183-205.
- 139. Manne S, Markowitz A, Winawer S, et al. Understanding intention to undergo colonoscopy among intermediaterisk siblings of colorectal cancer patients: A test of a mediational model. *Prev Med.* 2003;36(1):71-84.
- 140. Manne S, Markowitz A, Winawer S, et al. Correlates of colorectal cancer screening compliance and stage of adoption among siblings of individuals with early onset colorectal cancer. *Health psychology : official journal of the Division of Health Psychology, American Psychological Association*. 2002;21(1):3-15.
- 141. Gil AG, Wagner EF, Vega WA. Acculturation, Familism, and Alcohol use among Latino Adolescent Males: Longitudinal Relations. *Journal of Community Psychology*. 2000;28(4):443-458.
- 142. Kobayashi LC, Smith SG. Cancer Fatalism, Literacy, and Cancer Information Seeking in the American Public. *Health Educ Behav.* 2015.
- 143. Niederdeppe J, Levy AG. Fatalistic Beliefs about Cancer Prevention and Three Prevention Behaviors. *Cancer Epidem Biomar*. 2007;16(5):998-1003.
- 144. Shea JA, Micco E, Dean LT, McMurphy S, Schwartz JS, Armstrong K. Development of a Revised Health Care System Distrust Scale. *J Gen Intern Med.* 2008;23(6):727-732.
- 145. Boonyasiriwat W, Hung M, Hon SD, et al. Intention to undergo colonoscopy screening among relatives of colorectal cancer cases: a theory-based model. *Ann Behav Med.* 2014;47(3):280-291.
- 146. Lerman C, Daly M, Sands C, et al. Mammography Adherence and Pyschological Distress Among Women at Risk for Breast Cancer. *Journal of the National Cancer Institute*. 1993;85(13):1074-1080.
- 147. Fagerlin A, Zikmund-Fisher BJ, Ubel PA, Jankovic A, Derry HA, Smith DM. Measuring Numeracy without a Math Test: Development of the Subjective Numeracy Scale. *Med Decis Making*. 2007;27:672-680.
- 148. McNaughton CD, Cavanaugh KL, Kripalani S, Rothman RL, Wallston KA. Validation of a Short, 3-Item Version of the Subjective Numeracy Scale. *Med Decis Making*. 2015;35(8):932-936.
- 149. Parrott R, Silk K, Krieger JR, Harris T, Condit C. Behavioral Health Outcomes Associated with Religious Faith and Media Exposure about Human Genetics. *Health Communication*. 2004;16(1):29-45.
- 150. Kaphingst KA, McBride CM, Wade C, Alford SH, Brody LC, Baxevanis AD. Consumers' Use of Web-Based Information and their Decisions about Multiplex Genetic Susceptibility Testing. *Journal of Medical Internet Research*. 2010;12(3):e41.
- 151. Carere DA, Kraft P, Kaphingst KA, Roberts JS, Green RC. Consumers report lower confidence in their genetics knowledge following direct-to-consumer personal genomic testing. *Genetics in Medicine*. 2016;18(1):65-72.
- 152. Sheppard VB, Mays D, LaVeist T, Tercyak KP. Medical Mistrust Influences Black Women's Level of Engagement in BRCA1/2 Genetic Counseling and Testing. *Journal of the National Medical Association*. 2013;105(1):17-22.
- 153. Légaré F, Kearing S, Clay K, et al. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. *Can Fam Physician*. 2010;56(8):e308-314.
- 154. O'Connor AM. User Manual Decisional Conflict Scale. 1993; <a href="http://decisionaid.ohri.ca/docs/develop/User Manuals/UM Decisional Conflict.pdf">http://decisionaid.ohri.ca/docs/develop/User Manuals/UM Decisional Conflict.pdf</a>. Accessed January 19 2016.

PI Name: Kinney

Protocol Title: GRACE Project



- 155. Halbert CH, Kessler L, Collier A, et al. Low rates of African American participation in genetic counseling and testing for BRCA1/2 mutations: racial disparities or just a difference? *Journal of genetic counseling*. 2012;21(5):676-683.
- 156. Holmes-Rovner M, Kroll J, Schmitt N, et al. Patient satisfaction with health care decisions: the satisfaction with decision scale. *Med Decis Making*. 1996;16(1):58-64.
- 157. Wills CE, Holmes-Rovner M. Preliminary Validation of the Satisfaction with Decision Scale with Depressed Primary Care Patients. *Health Expectations*. 2003;6(2):149-159.
- 158. Brehaut JC, O'Connor AM, Wood TJ, et al. Validation of a decision regret scale. *Med Decis Making*. 2003;23(4):281-292.
- 159. Scherr CL, Christie J, Vadaparampil ST. Breast Cancer Survivors' Knowledge of Hereditary Breast and Ovarian Cancer following Genetic Counseling: An Exploration of General and Survivor-Specific Knowledge Items. *Public health genomics*. 2016;19:1-10.
- 160. Lerman C, Narod S, Schulman K, et al. BRCA1 testing in families with hereditary breast-ovarian cancer. A prospective study of patient decision making and outcomes. *Jama-J Am Med Assoc.* 1996;275(24):1885-1892.
- 161. Chew LD, Griffin JM, Partin MR, et al. Validation of screening questions for limited health literacy in a large VA outpatient population. *J Gen Intern Med.* 2008;23(5):561-566.
- 162. Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. *Family medicine*. 2004;36(8):588-594.
- 163. Hay JL, Shuk E, Cruz G, Ostroff JS. Thinking through Cancer Risk: Characterizing Smokers' Process of Risk Determination. *Qualitative Health Research*. 2005;15(8):1074-1085.
- 164. Hay JL, Primavera L, Gurmankin LA, Shuk E, Ostroff JS. Development and Validation of a Scale Assessing Novel Cancer-Related Risk Perceptions [Abstract]. *Society for Behavioral Medicine*. 2006;31:S190.
- 165. Jensen JD, Bernat JK, Davis LA, Yale R. Dispositional cancer worry: convergent, divergent, and predictive validity of existing scales. *Journal of psychosocial oncology*. 2010;28(5):470-489.
- 166. McCaul KD, Goetz PW. Worry. A paper on the National Cancer Institute website. http://dccps.nci.nih.gov/BRP/constructs/worry/index.html. Accessed January 19, 2016.
- 167. Derogatis LR. *BSI 18 Brief Symptom Inventory 18: Administration, Scoring, and Procedures Manual.* Minneapolis, MN: NCS Pearson, Inc; 2000.
- 168. Derogatis LR, Melisaratos N. The Brief Symptom Inventory: An Introductory Report. *Psychological Medicine*. 1983;13:595-605.
- Tabora J, BrintzenhofeSzoc K, Jacobsen P, et al. A New Psychosocial Screening Instrument for Use with Cancer Patients. *Psychosomatics*. 2001;42(3):241-246.
- 170. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. *J Health Soc Behav.* 1983;24(4):385-396.
- 171. Karam F, Be'rard A, Sheehy O, et al. Reliability and Validity of the 4-Item Perceived Stress Scale Among Pregnant Women: Results from the OTIS Antidepressants Study. *Research in Nursing and Health*. 2012;35:363-375.
- 172. Witte K. Fear Control and Danger Control: A Test of the Extended Parallel Process Model. *Commun Monogr.* 1994;61:113-134.
- 173. Birmingham WC, Hung M, Boonyasiriwat W, et al. Effectiveness of the extended parallel process model in promoting colorectal cancer screening. *Psycho-Oncology*. 2015;24(10):1265-1278.
- 174. Brug J, Steenhuis I, van Assema P, de Vries H. The Impact of a Computer-Tailored Nutrition Intervention. *Prev Med.* 1996;25:236-242.
- 175. Lipkus IM, Rimer BK, Halabi S, Strigo TS. Can tailored interventions increase mammography use among HMO women? *American Journal of Preventive Medicine*. 2000;18(1):1-10.
- 176. Street Jr RL. Physicians' Communication and Parents' Evaluations of Pediatric Consulations. *Med Care.* 1991;29(11):1146-1152.

PI Name: Kinney

Protocol Title: GRACE Project



- 177. Statistics USBoL. Overview of BLS Wage Data by Area and Occupation. 2016; <a href="http://www.bls.gov/bls/blswage.htm">http://www.bls.gov/bls/blswage.htm</a>. Accessed January 27, 2016.
- 178. Chang Y, Near AM, Butler KM, et al. Economic Evaluation Alongside a Clinical Trial of Telephone Versus In-person Genetic Counseling for BRCA1/2 Mutations in Geographically Underserved Areas. *Journal of Oncology Practice*. 2016;12(1):e1-e13.
- 179. Schwartz MD, Valdimarsdottir HB, Peshkin BN, et al. Randomized noninferiority trial of telephone versus inperson genetic counseling for hereditary breast and ovarian cancer. 2014;32(7):618-626.
- 180. Audrain J, Schwartz MD, Lerman C, Hughes C, Peshkin BN, Biesecker BB. Psychological Distress in Women Seeking Genetic Counseling for Breast-Ovarian Cancer Risk: The Contributions of Personality and Appraisal. *Ann Behav Med.* 1997;19(4):370-377.
- 181. Levy AG, Shea J, Williams SV, Quistberg A, Armstrong K. Measuring Perceptions of Breast Cancer Risk. *Cancer epidemiology, biomarkers & prevention : a publication of the American Association for Cancer Research, cosponsored by the American Society of Preventive Oncology.* 2006;15(10):1893-1898.
- 182. Witte K, Meyer G, Martell D. The Risk Behavior Diagnosis Scale. In: *Effective Health Risk Messages: A Step-by-Step Guide*. Thousand Oaks, CA: Sage Publications; 2001:67-76.
- 183. Cheah WH. Issue Involvement, Message Appeal, and Gonorrhea: Risk Perceptions in the US, England, Malaysia, and Singapore. *Asian Journal of Communication*. 2006;16(3):293-314.
- 184. Gil AG, Vega WA. Two different worlds: Acculturation stress and adaptation among Cuban and Nicaraguan families. *Journal of Social and Personal Relationships*. 1996;13:435-456.
- 185. Gil AG, Vega WA, Dimas J. Acculturative stress and personal adjustment among Hispanic adolescents. *Journal of Community Psychology.* 1994;22:43-54.
- 186. Rubin DB. Multiple Imputation for Nonresponse in Surveys In. New York: J. Wiley & Sons; 1987.
- 187. Holm S. A simple sequentially rejective multiple test procedure. *Scand J Stat.* 1979;6(2):65-70.
- 188. Kline RB. *Principles and Practice of Structural Equation Modeling*. Third ed. New York, NY: The Guilford Press; 2011.
- 189. Drummond M. *Methods for the economic evaluation of health care programmes*. New York, NY: Oxford University Press; 2015.
- 190. Gold MR, Patrick DL, Torrance GW, al. E. Identifying and valuing outcomes. In: Gold MR, Russel LB, Seigel JE, Weinstein MC, eds. *Cost-Effectiveness in Health and Medicine*. New York, NY: Oxford University Press; 1996:82-123.
- 191. Briggs AH, O'Brien BJ, Blackhouse G. Thinking outside the box: recent advances in the analysis and presentation of uncertainty in cost-effectiveness studies. *Annual review of public health*. 2002;23(1):377-401.
- 192. Fenwick E, O'Brien BJ, Briggs A. Cost-effectiveness acceptability curves--facts, fallacies and frequently asked questions. *Health economics*. 2004;13(5):405-415.
- 193. Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. *Health Educ Res.* 2006;21(5):688-694.
- 194. Harden SM, Gaglio B, Shoup JA, et al. Fidelity to and comparative results across behavioral interventions evaluated through the RE-AIM framework: a systematic review. *Systematic reviews*. 2015;4:155.
- 195. Glasgow RE, Askew S, Purcell P, et al. Use of RE-AIM to Address Health Inequities: Application in a low-income community health center based weight loss and hypertension self-management program. *Transl Behav Med.* 2013;3(2):200-210.
- 196. Patton MQ. *Qualitative research & evaluation methods : integrating theory and practice.* Fourth edition. ed. Thousand Oaks, California: SAGE Publications, Inc.; 2015.
- 197. Lwanga SK, Lemeshow S. *Sample size determination in health studies: A Practical Manual.* Geneva: World Health Organization; 1991.

PI Name: Kinney

Protocol Title: GRACE Project



198. PASS 13, NCSS, LLC, Kaysville, Utah, USA [computer program].